Protocol Title: Role of glare and spectral filtering on contrast sensitivity: A pilot study

Protocol CR-6501

Version: 4.0

Date: 02 November 2022

Investigational Products: None.

Keywords: Sphere platform, senofilcon A with a new UV/HEV filter (ACUVUE OASYS MAX 1-Day), senofilcon A without the new UV/HEV filter (ACUVUE OASYS 1-Day), daily wear, daily disposable, non-dispensing, contrast sensitivity function under photopic and mesopic conditions.

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This clinical trial will be conducted in compliance with ISO 14155:2020 Clinical investigation of medical devices for human subjects - Good clinical practice, and the Declaration of Helsinki.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| INTRODUCTION AND BACKGROUND | |
|---|---|
| <ol> <li>INTRODUCTION AND BACKGROUND</li></ol> | |
| <ol> <li>INTRODUCTION AND BACKGROUND</li></ol> | |
| <ol> <li>INTRODUCTION AND BACKGROUND</li></ol> | |
| INTRODUCTION AND BACKGROUND 1.1. Name and Descriptions of Investigational Products 1.2. Intended Use of Investigational Products 1.3. Summary of Findings from Nonclinical Studies 1.4. Summary of Known Risks and Benefits to Human Subjects | |
| | 25 |
| CHANGE HISTORY SYNOPSIS COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFI | DEFINITIONS OF TERMS |

| 6.3. Administration of Test Articles | 33 |
|---|---|
| 6.4. Packaging and Labeling | 33 |
| 6.5. Storage Conditions | 34 |
| 6.6. Collection and Storage of Samples | 34 |
| 6.7. Accountability of Test Articles | 34 |
| 7. STUDY EVALUATIONS | 35 |
| 7.1. Time and Event Schedule | 35 |
| 7.2. Detailed Study Procedures | 36 |
| VISIT 1 | 36 |
| FINAL EVALUATION | 45 |
| 7.3. Unscheduled Visits | 45 |
| 7.4. Laboratory Procedures | 47 |
| 8. SUBJECTS COMPLETION/WITHDRAWAL | 47 |
| 8.1. Completion Criteria | 47 |
| 8.2. Withdrawal/Discontinuation from the Study | 47 |
| 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 48 |
| 9.1. Systemic Medications | 48 |
| 10. DEVIATIONS FROM THE PROTOCOL | 49 |
| 11. STUDY TERMINATION | 50 |
| 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 51 |
| 13. ADVERSE EVENTS | 52 |
| 13.1. Definitions and Classifications | 52 |
| 13.2. Assessing Adverse Events | 54 |
| 13.2.1. Causality Assessment | 55 |
| 13.2.2. Severity Assessment | 55 |
| 13.3. Documentation and Follow-Up of Adverse Events | 55 |
| 13.4. Reporting Adverse Events | 57 |
| 13.4.1. Reporting Adverse Events to Sponsor | 57 |
| 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health A | |
| 13.5. Event of Special Interest | |
| 13.6. Reporting of Pregnancy | 58 |
| Johnson & Johnson Vision Care, Inc. | |
| 14. STATISTICAL METHODS | 59 |
| 14.1. General Considerations | 59 |
| 14.2. Sample Size Justification | 59 |

| 14.3. | Analysis Populations | 59 |
|---|---|---|
| 14.4. | Level of Statistical Significance | 60 |
| 14.5. | Primary Analysis | 60 |
| 14.6. | Secondary Analyses | 60 |
| 14.7. | Other Exploratory Analysis | 60 |
| 14.8. | Interim Analysis | 61 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 61 |
| 14.10 | . Procedure for Reporting Deviations from Statistical Plan | 61 |
| 15. DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 61 |
| 15.1. | Electronic Case Report Form/Data Collection | 61 |
| 15.2. | Subject Record | 62 |
| 15.3. | Trial Registration on ClinicalTrials.gov | 62 |
| 16. DA | TA MANAGEMENT | 62 |
| 16.1. | Access to Source Data/Document | 62 |
| 16.2. | Confidentiality of Information | 62 |
| 16.3. | Data Quality Assurance | 63 |
| 16.4. | Data Monitoring Committee (DMC) | 63 |
| 17. CL | INICAL MONITORING | 63 |
| 18. ET | HICAL AND REGULATORY ASPECTS | 64 |
| 18.1. | Study-Specific Design Considerations | 64 |
| 18.2. | Investigator Responsibility | 64 |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 64 |
| 18.4. | Informed Consent | 65 |
| 18.5. | Privacy of Personal Data | 66 |
| 19. ST | UDY RECORD RETENTION | 67 |
| 20. FIN | NANCIAL CONSIDERATIONS | 68 |
| 21. PU | BLICATION | 68 |
| 22. RE | FERENCES | 68 |
| APPEN | DIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES | ) 70 |
| APPEN | DIX B: PATIENT INSTRUCTION GUIDE | 71 |
| APPEN | DIX C: PACKAGE INSERT (APPROVED PRODUCT) | 72 |
| APPEN | DIX D: | 122 |
| _ | LENS FITTING CHARACTERISTICS | |
| _ | SUBJECT REPORTED OCULAR SYMPTOMS | |
| _ | DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRAC | |

### PROTOCOL TITLE, NUMBER, VERSION AND DATE

Title: Protocol Title: Role of glare and spectral filtering on contrast sensitivity: A pilot study

Protocol Nmnber: CR-6501

Version: 4.0

Date: 02 November 2022

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JNC) 7500 Centurion PaJkway Jacksonville, FL 32256

#### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail or telephone within 24 hoursofl earning of a Serious AdverseEvent. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessaly assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatoly requirements and applicable U.S. federal regulations,<sup>3</sup> ISO 14155:2020,<sup>1</sup> and the Declaration of Helsinki.<sup>2</sup>



| Approver | See Electronic Signature Report | |
|----------|---------------------------------|------|
| | | DATE |

### **CHANGE IDSTORY**

| Version | Originator | Description of Change(s) | Justification | Date |
|---|---|---|---|---|
| | | and Section Number(s)<br>Affected | for Change | |
| I.O | | Original Protocol | N/A | 21 September 2022 |
| 2.0 | | Updated Section 5.1 Test Alticle Allocation to clarify that there will be only one lens assignment for the two light sources (i.e., without glare and with olare er sub ect | To align the randomization plan with study procedures | 04 October 2022 |
| 3.0 | | 1. Section 7.2 - VI Step<br>1.21, 1.22, 1.24 and 1.25,<br>changed spatial frequency<br>2.3 to 3.2 to match lens<br>fitting schedule. | 1. Accuracy | 24 October 2022 |
| | | 2. Section 1.5 - changed "to believe that" to "for why" / changed "obtainable" to "of interest" | 2. Per Legal<br>TeamReview | |
| 4.0 | | Section 7.2 Steps 1.21,<br>1.22, 1.24 and 1.25,<br>updated area under the<br>contrast sensitivity curve<br>range from 100 to 5.00 | Accuracy | 02 November 2022 |

### **SYNOPSIS**

| Protocol Title | Protocol Title: Role of glare and spectral filtering on contrast sensitivity: A pilot study |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Clinical trial phase: Feasibility Design control phase: Phase 3 |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the Sponsor |
| Test Article(s) | Investigational Products: None. Approved Products: 1. senofilcon A with a new UV/HEV filter (ACUVUE OASYS MAX 1-Day). 2. senofilcon A without a new UV/HEV filter (ACUVUE OASYS 1-Day). |
| Wear and Replacement<br>Schedules | Wear Schedule: daily wear Replacement Schedule: daily disposable |
| Objectives | The purpose of this study is to evaluate the role of a test lens on contrast sensitivity with and without glare. Primary Objectives: The primary objective is to evaluate the visual performance characteristics of a new UV/HEV filter under conditions of an HEV-rich ecologically-valid light source. |

| C. 1 F. 1 | D: D 1 : (() |
|---|---|
| Study Endpoints | Primary Endpoint(s) |
| | • Area under the curve of photopic contrast sensitivity function under bright light conditions (approx. 120 cd/m2) with a broadband glare source. |
| | Secondary Endpoint(s) |
| | • Area under the curve of mesopic contrast sensitivity under dim light conditions (approx. 3 cd/m2) with a broadband glare source. |
| | Other Observations: |
| | <ul> <li>Area under the curve of photopic contrast sensitivity function under bright light conditions (approx. 120 cd/m2) without a broadband glare source.</li> <li>Area under the curve of mesopic contrast sensitivity under dim light conditions (approx. 3 cd/m2) without a broadband glare source.</li> </ul> |
| Study Design | This is a split-plot design with two parallel arms consisting of randomized photopic and mesopic conditions where subjects are also randomized contralaterally to the Test and Control lenses within each arm. This study will be non-dispensing, controlled, and double-masked. Subjects will be assigned randomly to the photopic or the mesopic condition arm. Each subject will be fitted with a Test lens on one eye and a Control lens on the other eye within each condition arm. The randomization will be stratified by age with a 1:1 ratio for the two age ranges (18-40 years; 41-65 years). |
| | There will be a total of 1 visit: |
| | • Visit 1: Screening, baseline evaluation and lens fit #1 and #2. Evaluation of lens 1 and 2. Final evaluation. |
| | See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). |
| Sample Size | Approximately 44 subjects will be enrolled with the intent to complete approximately 20 in each group (photopic and mesopic). |
| Study Duration | This study is non-dispensing and is completed in a single visit. The enrollment period is approximately 2 months. |

| Anticipated Study<br>Population | Subjects must be habitual wearers of silicone hydrogel contact lenses worn on a daily wear basis. Subjects can be of any gender, race, and ethnicity that meet the eligibility criteria. |
|---|---|
| Eligibility Criteria -<br>Inclusion | Potential subjects must satisfy all of the following criteria to be enrolled in the study: |
| | Inclusion Criteria following Screening |
| | The subject must: |
| | <ol> <li>Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Be between 18 and 65 (inclusive) years of age at the time of screening.</li> <li>By self-report, habitually wear spherical silicone hydrogel soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.</li> <li>Possess a wearable pair of spectacles that provide correction for distance vision.</li> </ol> |
| | Inclusion Criteria at Baseline Evaluation |
| | <ul> <li>6. The spherical equivalent of the subject's vertex corrected distance refraction must be between -1.00 D and -6.00 D (inclusive) in each eye.</li> <li>7. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be between 0.00 D and 1.00 D (inclusive) in each eye.</li> <li>8. The best corrected, monocular, distance visual acuity must be 20/25 or better in each eye.</li> </ul> |

# Eligibility Criteria - Exclusion

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening

The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Be currently using any ocular medications or have any ocular infection of any type.
- 3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjogren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
- 4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
- 5. Be currently wearing monovision or multifocal contact lenses.
- 6. Be currently wearing lenses in an extended wear modality.
- 7. Have participated in a contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 8. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.

Exclusion Criteria at Baseline Evaluation

The subject must not:

9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including

| | entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis). 10. Have a history of strabismus or amblyopia. 11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions. 12. Have had any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.). 13. Have signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar). 14. Have a history of eyelid injury, surgery or procedure that resulted in abnormal eyelid position or movement. |
|---|---|
| Disallowed Medications/Interventions | Subjects taking and ocular medications will not be allowed to participate. See section 9.1 for details regarding disallowed systemic medications. |
| Measurements and Procedures | All measurements will be taken with and without an ecologically-valid glare source. Approximately half of the subjects will be tested under photopic conditions and the other half under mesopic conditions. |
| Microbiology or Other<br>Laboratory Testing | None. |
| Study Termination | The occurrence of an Unanticipated Adverse Device Effect (UADE) or Serious Adverse Event (SAE) for which a causal relationship to a test article cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | An ecologically-valid broadband glare source that emulates natural sunlight in spectral content across the visible spectrum will be used. RevitaLens will be used to return any problematic lenses to the Sponsor. |

| and Study | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |
|---|---|
| Institution(s)/Site(s) | included in the study I rial Master File. |

Figure 1:Study Flowchart



C R -6 501, v -4.0

# COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADE Adverse Device Effect

ADHD Attention Deficit Hyperactivity Disorder
AE Adverse Event/Adverse Experience
BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience
COM Clinical Operations Manager
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure

ICH The International Council for Harmonization

IEC Independent Ethics Committee IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc. LASIK Laser-Assisted in Situ Keratomileusis

OD Right Eye
OS Left Eye
OU Both Eyes

PIG Patient Instruction Guide
PQC Product Quality Complaint
PRK Photorefractive Keratectomy
PRO Patient Reported Outcome

QA Quality Assurance

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Contrast sensitivity functions (CSF) have wide scientific and clinical use (NRC, 1985). Their value, however, depends critically on their reliability and their ecological validity. In most vision experiments, CSFs are measured with a CRT oscilloscope or computer monitor (or even less precisely, with wall charts like the Peli-Robson or the CSV-1000), which allows relatively simple electronic control of both spatial frequency and contrast. A common method, for example, of measuring CSF is employed by the Metropsis system (Cambridge Research). This system presents a series of sine-waves (as Gabor patches) on a highly calibrated monitor with computer control over presentations and refined psychophysical procedures (the modern version of the original method used on a CRT screen by Campbell and Robson, 1968). The Metropsis system has been used to evaluate spatial vision issues in a variety of patient populations (e.g. to assess the effects of brain injury, smoking or toxic exposures; Nguyen et al., 2017; Costa et al., 2012; Fernandes et al., 2017).

Fernandes et al. (2019) evaluated the Metropsis method on 55 normal subjects. The curves provided by Fernandes were unusually flat (e.g., between about 0.2-8.8 cycles/degrees; shown in Figure 2) with intraclass correlations of around 0.71 when testing 20 subjects (the authors note that this is considerably higher than intraclass correlations generated by the CSV-1000 (0.19), Pelli-Robson (0.18), Vistech FDT (0.36) or Miller=Nadler (0.36) CSF tests.

Figure 2: Binocular contrast sensitivity values derived from Figure 2 of Fernandes et al. (black line and symbols) compared to data from Scheiber et al (red line and symbols: 20 year-old observers). Note the deviation at the lower frequencies.



Reliability is, of course, critical in a prognostic device. As originally expressed by the National Research Council (1985), "The value of the contrast sensitivity function in predicting performance on complex visual tasks and in discriminating among individuals in their ability on these tasks needs to be further explored." If the amount of variance explained (r2) is only 50% (meaning a measure predicts half of the variance in that same measure taken at a different time), then its ability to predict other variables is, perforce, less than 50%. It would be optimal to have a system for measuring CSF that has better reliability.

The other major issue with CSF curves measured using monitors is their inconsistency across studies (convergent validity). A classic curve in the CSF literature, for example, comes from van Nes and Bouman (1967) shown below (Figure 3).

Figure 3: CSF data from van Nes and Bouman. Note that the peak sensitivity value is near around 5 cyc/deg and sensitivity is peaking around 400-500 (about twice the peak from the Metropsis sample shown in Fig 2). (also note the similarity in the curves across luminance-from 90-900 trolands, analogous to 3 to 300 cd/m<sup>2</sup> based on a 2 mm pupil).



The shape of the curve is similar to the classic curve reported by Campbell and Robson (1968). The peak is quite different (3 cycles/degree, contrast sensitivity = 700). Shown in Figure 4.

Figure 4: CSF according to Campbell and Robson (1968).



Contrast these peaks with others often reported in the literature. Here, for example, is a sample of young and older subjects from Elliott et al. 2009 (Figure 5).

Figure 5: Figure from Elliott et al. (2009); data are from older (red) and younger (black) subjects with various abe1rntions co1Tected. In this study the peak is around 8 cycles per degree and contra.st sensitivity is about 80.



If one does a wide survey of nonnal CSF curves in the literature, you can find wide divergence in the shape of CSF curves and in peak sensitivity (a range by at least a factor of ten). One reason is lack of standardizing many of the variables that drive the curves (size, illuminance, etc), although even when this is done, convergent validity seems to be poor (Buhren et al., 2006). Another reason is that the modulation depth of the stimuli are ra.rely directly calibra.ted (on monitors, the actual values are derived not actually measured in place). This is a particular issue with CRTs (Garcia-Perez and Peli, 2001). The quality of the stimulus display ranges from paper wall charts (e.g., Peli-Robson) to cathode-ra.y tubes to various types of monitor designs (e.g., Metropsis). The range of procedures also varies from deriving tlu esholds from relatively long psychometric functions (like in Metropsis) to vely rough approximations (e.g., CSV-1000), see Figure 6).


Figure 6: The stimuli used in the CSV-1000 test (right side shows the glare condition).





This lack of standardization is likely why CSF methods often have poor predictability and ecological validity. This was originally tested by Owsley and Sloane (1987):

"A major assumption underlying the use of contrast sensitivity testing is that it predicts whether a patient has difficulty seeing objects encountered in everyday life. However, there has been no large-scale attempt to evaluate whether this putative relationship actually exists."

Owsley and Sloane measured Snellen acuity and the CSF of 93 subjects (aged 20-77 yrs.). These measures were then compared with target images (faces, road signs, and other objects) that were placed on back-illuminated slides. These slides were placed in an optical system that allowed the contrast within the object to be varied. These authors found that Snellen acuity did not predict threshold identification of these "real-world targets." CSF did predict real-world performance but explained only 25-40% of the variance. This supports the potential utility of CSF as a measure of vision in everyday life while also highlighting a potential opportunity to develop new methods of measuring CSF to improve its ability to predict vision in everyday life.

Fortunately, high quality sine-wave transparencies are available from Applied Image, who can custom make the sine-waves and calibrate them precisely. These targets have low harmonic distortions (2% or less) and are available cemented between large (100 x100 in) squares of glass. They are nearly spectrally flat. These were originally used in a study by Hammond et al. (2012) and Fletcher et al. (2014). These foundational studies showed that CSF can be measured using real optics and carefully controlled and calibrated conditions.

Another challenge when measuring CSF is to introduce the kind of stressors that actually affect spatial vision in the real world. One such stressor is glare. The primary source of glare in the

real world is the sun (Mitra, 2014, Sun et al., 2018). A major issue with many of the existing glare systems (see Figure 5) is that the glare source that is used does not resemble actual sunlight (Tungsten-Halogen is a common source, the Metropsis uses white LEDs). In our study we will use white light with xenon as the source and filtered to precisely match specific phases of sunlight. Another important consideration is the angle. Often glare sources are made to surround the entire display. For example, the CSV-1000 mounts the glare source on the sides, Metropsis mounts the glare source vertically as shown in Figure 7.

Figure 7: The glare source of the Metropsis is based on white LEDs mounted vertically.



In the real world, the glare source (say the sun) and the visual target (say a stop sign) are relatively far away. In some instances, this distance homogenizes the light scatter interfering with perception of the stimulus. In a clinic, the stimulus and glare source are only a few feet away making the glare less uniform (it is more intense as it gets closer to the source). To optimally emulate real world visual conditions, the veiling light should be relatively homogenous.

#### Issues revealed by our previous pilot study:

In our previous pilot study, we measured CSF (photopic and mesopic) under regular and glare conditions. This was done to assess whether CSF with our HEV-absorbing test lens differed from a clear control. Although preliminary testing demonstrated a significant reduction in CSF with glare, in a second cohort, we found that our glare condition did not reduce CSF (i.e. the CSF curves were the same in the glare and non-glare condition). Hence, the HEV test lens did not have a reduction to correct. Why did our glare condition not work?

In our previous discussion we argued that the measures of CSF provided by the Metropsis were highly variable, likely reducing our ability to discriminate small differences between the two test conditions. Another possible methodological limitation might have been the positioning of the glare source. One possible reason why the glare condition did not reduce the CSF was

that it was insufficiently homogeneous and too far from the line of sight. Like in real life, people will reflexively try to see around glare (dive1t their eyes to the least glaring portion of the image) and this may have been possible with our glare ring a1Tangement (the preliminruy testing was sho1t and composed of subjects that were highly compliant). In order to really test the effects of glru·e, the glare source needs to be perfectly homogeneous and made such that it cannot be avoided. Our current study is designed to address both the reliability issues with Metropsis and the homogeneity of the glare source.

### University of Georgia contrast sensitivity testing apparatus:

The simplified design of this system was based on many of the satne principles that were worked out on the much more elaborate optical systems used in Hammond et al. (2012) and Fletcher et al. (2014). A custom-built apparatus was used to measure contrast sensitivity functions at 1.6, 3.2, 8, 16 and 24 cycles/degree (See the schematic in Figure 8).

Figure 8: University of Georgia CSF Apparatus



The system uses two green (520 nm) lasers (Ll and L2) that are spatially diffused using two six-inch circulru integrating spheres (aluminum hemispheres painted on the interior with highly diffusing, 98% reflecting, non-luminescent, white paint, Labsphere, N01th Sutton, NH). To measure contrast sensitivity, the intensity of the light source (Ll and L2) is independently adjusted using circular neutral density wedges (Wl and W2). The two spheres pass the homogeneous green light through two exit poris (~3.5 deg circular). The green laser light source is positioned with respect to the surface of the integrating sphere in such a way as to create a completely homogeneous light at the plane of the retina, essentially a Lambertian

CR-6501, v 4.0

emitter. This creates a visual stimulus with luminance that is relatively independent of exact eye position.

Light from Sphere 1 passes through a 2-inch diameter sine wave grating (1.6, 3.2, 8, 16, or 24 cyc/deg based on a distance of 36 inches to the plane of the eye). These gratings are placed in a mount that can be rotated to the left or right (15 degree cant) in order to provide a forced choice procedure. A thin optomechanical shutter (Thor Labs) by L1 allows the intermittent exposure (-1 second exposures) of the grating stimulus. Light from Sphere 2 combines with Sphere 1 and wedge adjustment allows for constant variation in the modulation of the sine waves. A dedicated photodetector (Graseby Optronics United Detection Technology (UDT) with a photometric lens Orlando, FL) is used to constantly monitor the luminance output (half of the combined beam going to the detector and half going to the eye of the subject to maintain a constant luminance of 65 cd/m2). The gratings were calibrated by the manufacturer and confirmed within the system by moving a tiny pinhole aperture (-1/2 mm) and photodetector (ILT 950, International Light Technologies, Peabody MA) across and very close to the surface of the grating while changing the position of the wedges. Optical baffling was used throughout (not shown in the schematic) to prevent light noise between the channels.

Subject head position is maintained using a forehead and chin rest assembly (36 inches from the grating). Contrast thresholds are calculated based on the Michelson contrast formulation. A method of limits is used to obtain threshold (ascending and descending). A method of constant stimuli combined with the forced choice procedure (canted left or right) is used to refine the threshold determination to approximately 75% correct (based on 10 determinations).

To measure CSF, two ascending and two descending thresholds will be taken for each grating, with grating order randomly assigned for each participant. If raw values vary by more than 200 arbitrary units on the wedge display, the forced choice / constant stimuli method will be used to arrive at a more exact threshold.

#### Glare system

The glare system is composed of a one-channel optical system with a 1000-watt xenon light source. Light exits the housing and is collimated using an achromatic plano-convex lens. This collimated light passes through a water baffle (a clear tube with optical flats on either end) that removes heat without altering the light spectrum. The collimated light passes through a series of achromatic plano-convex lenses that alternately focus and collimate the light. A color correcting filter (e.g., Daylight Blue Filter, Edmunds Optics) will be used to achieve a CCT of at least 6500K. The collimating light will be approximately three inches in diameter. The entire system is orthogonal to the CSF device. At the junction between the exit port of the CSF device a large thin glass beam-splitter (analogous to a large cover slip) will be used. This creates a large perfectly homogeneous glare source between and co-liner with the grating and the eye of the subject. See Figure 9.

Figure 9: University of Georgia glare system



### 1.1. Name and Descriptions of Investigational Products

This study will evaluate two (2) senofilcon A designs with and without a new UV/HEV filter. The Test lens is FDA-approved and pending commercial distribution. The Control lens is ACUVUE OASYS 1-Day with HydraLuxe<sup>TM</sup> Technology. Further details about the test articles are found in section 6 of this protocol.

### 1.2. Intended Use of Investigational Products

The intended use of the investigational products is for correcting myopia (Test and Control) and improving visual performance characteristics under applicable conditions (Test). The study articles will be worn contralaterally in a daily wear, daily disposable modality for 1-2 hours.

### 1.3. Summary of Findings from Nonclinical Studies

Not Applicable - Marketed product only.

### 1.4. Summary of Known Risks and Benefits to Human Subjects

Benefits to the subjects include the correction of their refractive error with the potential of improved visual performance in HEV environments. The risks of wearing soft contact lenses are well known and are described in the Investigator's Brochure and Informed Consent. The material safety testing/lens release criteria was determined based on the Risk Assessment.

For the most comprehensive risk and benefit information regarding Test and Control lenses, refer to the latest version of the package insert.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

The new HEV-filter in the Test lens has been evaluated in two previous objective-based studies: and and an an an an an an an are an area. In both studies, psychophysical evaluations were carried out on an optical breadboard system using a broadband light source that emulated sunlight in spectral content. These studies demonstrate that benefits of a HEV-filter can be seen when tested in an HEV-rich environment such as natural sunlight:

- 1. (n=60 cohort): when compared to a similar contact lens without the new UV/HEV filter, the Test lens demonstrated statistical superiority in the following metrics:
  - o 2-point light threshold
  - Halo diameter
  - Starburst diameter
  - o Disability glare
  - Discomfort glare
  - Chromatic contrast
- 2. (n=58 cohort): when compared to a similar contact lens without the new UV/HEV filter (different control lens than statistical superiority in the following metrics:
  - o 2-point light threshold
  - Halo diameter
  - Discomfort glare
  - Chromatic contrast
  - Photostress recovery

To further, many of the metrics noted above provide a reason for why the specific hypotheses of this study are of interest. Mainly:

| 1. | Improved contrast | |
|---|---|---|
| | 0 | In and and , disability glare was measured by noting the intensity |
| | | of a broadband light source needed to obscure a central grating target. The results |
| | | from this study demonstrate that subjects can see a high contrast central grating |
| | | target under HEV-rich conditions such as sunlight better with an HEV-filter. |
| | 0 | In and and, heterochromatic contrast was measured by noting the |
| | | intensity of a 460 nm light source needed to obscure a 580 nm central grating |
| | | target. The results demonstrate an improved ability to detect edges while wearing |
| | | an HEV-filter. |
| _ | _ | |

2. Improved low light vision

o In and and proved, broadband light that emulated sunlight in spectral content was used to generate a point source of light. The halo and starburst

diameters of that light were measured using precision calipers. The results demonstrate that positive dysphotopsia, which is most prevalent in dim illumination, can be improved with an HEV-filter. <sup>4-6</sup>

(n=59) was a method development pilot study intended to test contrast sensitivity and resolution acuity under various conditions. The learnings from that study are mentioned throughout the introduction of this protocol and incorporated into the current study.

Refer to the Package Insert (Appendix C) for additional information about the study lenses.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

### 2.1. Objectives

The intent of this study is to determine whether or not the Test lens is likely to provide visual benefits under conditions for which it was designed. All mentions of broadband glare, or just glare, are referring to an ecologically-valid light source that emulates sunlight in spectral content.

### Primary Objective(s)

The primary objective is to evaluate the visual performance characteristics of a new UV/HEV filter under conditions where an ecologically-valid light source is present.

### 2.2. Endpoints

### Primary Endpoint(s)

• Area under the curve of photopic contrast sensitivity function under bright light conditions (~120 cd/m2) with a broadband glare source.

### Secondary Endpoint(s)

• Area under the curve of mesopic contrast sensitivity under dim light conditions (~3 cd/m2) with a broadband glare source.

#### Other Observations:

- Area under the curve of photopic contrast sensitivity function under bright light conditions (~120 cd/m2) without a broadband glare source.
- Area under the curve of mesopic contrast sensitivity under dim light conditions (~3 cd/m2) without a broadband glare source.

### 2.3. Hypotheses

#### Primary Hypothesis

No primary hypothesis will be tested. The primary endpoint will be descriptively summarized.

#### Secondary Hypothesis

No secondary hypothesis will be tested. The secondary endpoint will be descriptively summarized.

### **Exploratory Hypotheses**

- The Test lens will provide greater photopic contrast sensitivity compared to the Control lens under conditions of a broadband glare source.
- The Test lens will provide greater mesopic contrast sensitivity compared to the Control lens under conditions of a broadband glare source.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Subjects must be habitual wearers of silicone hydrogel contact lenses worn on a daily wear basis. Subjects can be of any gender, race, and ethnicity that meet the eligibility criteria.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

Inclusion Criteria following Screening

The subject must:

- 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Be between 18 and 65 (inclusive) years of age at the time of screening.
- 4. By self-report, habitually wear spherical silicone hydrogel soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
- 5. Possess a wearable pair of spectacles that provide correction for distance vision.

#### Inclusion Criteria at Baseline Evaluation

- 6. The spherical equivalent of the subject's vertex corrected distance refraction must be between -1.00 D and -6.00 D (inclusive) in each eye.
- 7. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be between 0.00 D and 1.00 D (inclusive) in each eye.
- 8. The best corrected, monocular, distance visual acuity must be 20/25 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening

The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Be currently using any ocular medications or have any ocular infection of any type.
- 3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjogren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
- 4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
- 5. Be currently wearing monovision or multifocal contact lenses.
- 6. Be currently wearing lenses in an extended wear modality.
- 7. Have participated in a contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 8. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.

### **Exclusion Criteria at Baseline Evaluation**

### The subject must not:

- 9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
- 10. Have a history of strabismus or amblyopia.
- 11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
- 12. Have had any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).
- 13. Have signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar).
- 14. Have a history of eyelid injury, surgery or procedure that resulted in abnormal eyelid position or movement.

### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

### 4.1. Description of Study Design

This is a split-plot design with two parallel arms consisting of randomized photopic and mesopic conditions where subjects are also randomized contralaterally to the Test and Control lenses within each arm. This study will be non-dispensing, controlled, and double-masked. The study lenses will be worn in a daily wear modality for 1-2 hours. Subjects will not have access to the study lenses at the conclusion of their visit.

### 4.2. Study Design Rationale

This is a split-plot design with two parallel arms consisting of randomized photopic and mesopic conditions where subjects are also randomized contralaterally to the Test and Control lenses within each arm. The photopic and mesopic conditions will be the two-parallel arms so that these two conditions can be assessed separately. There are several benefits to the choice of the contralateral design within each condition arm. First, a contralateral design will allow us to compare performance within the same individual, ostensibly with the same baseline light sensitivity by eye. Second, other subject factors that can influence visual performance, such as iris color and absorption of test lights via macular pigment, are better controlled using this design. Third, in psychophysical testing, which is the gold standard for many of the visual functions being tested, participants make judgments about some event threshold, such as when an image disappears. Participants may have different criteria for threshold events that are internally consistent within subjects but can vary between subjects. A contralateral design allows the investigational lens to be compared within subjects, with consistent criteria for threshold events.

#### 4.3. Enrollment Target and Study Duration

This study will have an enrollment target of 44 subjects, with a target of at least 40 to complete (approximately 20 subjects [10 subjects from the 18-40 years of age range; 10 subjects from the 41-65 years of age range] in each arm). The study will be conducted at a single clinical site. A subject will be considered enrolled upon signing of the informed consent form.

There will be 1 visit total per subject; total study duration including the enrollment period is expected to be approximately 2 months. If subjects discontinue prior to the final evaluation, then additional subjects may be enrolled at the discretion of the study sponsor to maintain the sample size plan. The investigation will end at the time that the study data is hard locked.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

### 5.1. Test Article Allocation

Use of the test articles will be randomized using a lens fitting schedule supplied by the study biostatistician. The randomization scheme will be generated by the unmasked biostatistician using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).<sup>7</sup> The clinical site will follow the lens fitting schedule

provided and will complete enrollment according to the randomization list and will not preselect or pre-assign subjects.

Randomly-permuted block randomization will be used to avoid bias in the assignment of subjects to treatment and to enhance the validity of statistical comparisons across treatment groups. Randomization will be stratified into two age groups (18-39 years old and 40-65 years old) using a 1:1 allocation ratio. Subjects will be first assigned randomly to the photopic or the mesopic condition arm. The order of the light sources within each condition arm is predetermined: visual performance will be assessed under the no broadband light source (without glare) condition first and then assessed under the broadband light source (with glare) condition. Within each condition arm, subjects will be randomized to either wear the Test lens in the left eye and the Control lens in the right eye or the Control lens in the left eye and the Test lens in the right eye. There will be only one lens assignment for the two light sources (i.e., without glare and with glare) per subject. Under each light source condition, the right eye will always be tested first. Once a participant's lens assignment has been randomized, the order of test stimuli will also be randomly assigned. Five spatial frequencies for contrast sensitivity testing (1.6, 3.2, 8, 16, and 24 cycles per degree) will be tested in the no-glare condition, and in the glare condition. Spatial frequency order will be randomized for both the no-glare condition and the glare condition for each subject eye.

Randomization will be performed at visit 1. The following must have occurred prior to randomization:

- Informed consent must have been obtained.
- The subject must have met all eligibility criteria.
- The subject's screening and baseline information must have been collected.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule to obtain the test article assignment for that subject prior to dispensing.
- 2. Investigator or designee will record the subject's number on the appropriate line of the lens fitting schedule.
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 5.2. Masking

This is a double-masked trial. Masking will be used to reduce potential bias. Subjects will be unaware of the identity of the investigational product assigned in the left eye and right eye. Investigators involved in the clinical assessment and data collection will be masked as to the identity of the investigational product. However, the clinician fitting the lenses may be aware of the identity of the investigational product due to the slight color difference between the

study lenses, and the clinician won't be involved in any clinical assessment or data collection of the study.

### 5.3. Procedures for Maintaining and Breaking the Masking

Evely attempt will be made to keep the clinical trial personnel involved in the study (e.g. data management, biostatistician and clinical operations) unaware of the identity of the assigned study lenses. The identity of the study lenses will be masked by having the blister packs labeled with the study number, lot number, sphere power, expiration date and the randomization codes. Only the urunasked biostatistician generating the lens fitting schedule will have access to the decode infonnation that allows matching of the randomization codes to the test aiiicles. The medical monitor will also have access to the decode info1mation in case breaking the mask is necessaly for the urgent medical treatment of a subject.

Under no1mal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Othe1wise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the sponsor must be info1med as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The investigator is also advised not to reveal the study treatment assignment to the clinical site or sponsor personnel.

If subjects discontinue prior to the final evaluation, then additional subjects may be emolled at the discretion of the study sponsor to maintain the sainple size plan.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Atiicles

| | Test | Control |
|-------------------------|---------------------|--------------------|
| Name | AOMAX | AOlD |
| Manufacturer | JNC | JNC |
| | | _ |
| Lens Matelial | senofilcon A C3 | senofilcon A C3 |
| Nomina1 Diameter | 8.5<br>14.3 | 8.5<br>14.3 |
| Nominal Distance Powers | -1.00 throu h -6.00 | -1.00 throuo -6.00 |
| Water Content (O tional | 38 | 38 |
| Center Thickness | 0.085 | 0.085 |
| Ox oen Pelmeabilit Dk | 103 | 103 |

| | Test | Control |
|--------------------------------------|--------|---------|
| Wear Schedule in Cunent Study | Daily | Daily |
| Replacement Frequency | Daily | Daily |
| Packaging Fonn (vial, blister, etc.) | Bhster | Bhster |
| New UV/HEV-blocker | Yes | No |

AOMAX = ACUVUE® OASYS MAX 1-Day, AOID = ACUVUE® OASYS 1-Day

Approximately 11 lenses per stock keeping unit (SKU) will be provided based on 44 subjects, I-period, contralateral, non-dispensing design, US population n01mahzed far peak SKUs.

## 6.2. Ancillary Supplies/Products

The fallowing solutions will be used in this study:

Table 2: Ancillaiy Supphes

| _ | Solutions | | | |
|---|---|---|---|---|
| Solution<br>Name/Description | Acuvue <sup>TM</sup> RevitaLens<br>Multipurpose Solution | Single use<br>Eye-Cept®<br>Rewetting<br>Drops | LacriPure<br>Sahne<br>Solution | ScleralFil Preservative Free Sahne Solution |
| Manufacturer | Johnson & Johnson<br>Vision | Optics<br>Laborato1y | Menicon | Bausch &<br>Lomb |
| Preservative | alexidine<br>dihydrochloride<br>0.00016% and<br>polyquatemium-1<br>0.0003% | None | None | None |

Lens cases and fluorescein strips (either 0.6 mg or 1.0 mg) will be supplied far use as needed.

#### 6.3. Administration of Test Articles

Test aiticles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set falth in this clinical protocol. Subjects will be dispensed an adequate supply of test aiticles to complete the study. Lost or damaged test aiticles may be replaced at the discretion of the investigator and/or the sponsor.

### 6.4 Pa ck aging and Labeling

The study aiticles will be packaged in blisters as the primary packaging. The study aiticle will be over-labeled to mask the subject and investigators to the identity of the lens. The study aiticles will be in plastic bags as the secondaly packaging folm. The samp le study label is shown below (Figure 10).


Figure 10: Packaging Labels



## 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

## **6.6.** Collection and Storage of Samples

No samples will be collected as part of the study procedures.

When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.

## 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test aiticles from the subjects at the end of the subject's paiticipation. Subject returned unused test aiticles must be sepai ated from the clinical study invent01y of un-dispensed test aiticles and must be labeled with the subject number and date of return. Following final reconciliation of test aiticles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately</u>.

#### 7. STUDYEVALUATIONS

### 7.1. Time and Event Schedule

Table 3: Time and Events

| | Visit 1 |
|---|---|
| Visit Information | <b>Screening, Baseline, Fitting</b> / |
| VISIT THIOT HIACION | Assessment |
| | Final Evaluation |
| Time Point | DayO |
| EstimatedVisit Dmation | 3.0 homs |
| Statement of Infonned Consent | Х |
| Demographics | X |
| Medica! Hist01y/Concomitan t Medications | X |
| Habitual Contact Lens Infolmation | X |
| Eligibility Following Screening | X |
| Entrance Visual Acuity | X |
| Subjective Sphero-Cylindrical Refraction and best- | X |
| colTected VA | |
| Eve Doininancy | X |
| Slit Lamo Bioinicroscoov | X |
| Eligibility Following Baseline Evaluation | X |
| Lens Selection | X |
| Lens Inselt ion & Settling | X |
| Visual Acuity and Over Refraction | X |
| Lens Power Modification (if applicable) | X |
| Subject Repolied Ocular Symptoms | X |
| Visual Acuity | X |
| General Fit Assessment | X |

| Visit Information | Visit 1 Screening, Baseline, Fitting / Assessment Final Evaluation |
|---|---|
| Time Point | DavO |
| Estimated Visit Duration | 3.0 hours |
| Vision Assessments: photopic and mesopic contrast sensitivity | X |
| Exit Snellen Distance Visual Acuity | X |
| Study Completion | X |

## 7.2. Detailed Study Procedures

### VISIT 1

The subjects must present to Visit 1 wearing spectacles, not having wom contact lenses on the day of the visit.

| | Visit 1: Screenin | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Infonned Consent | Each subject must read, understand, and sign the Statement of Infonned Consent before being emolled into the study. The Principal Investigator or his/her designee conducting the info1med consent discussion must also sign the consent f01m. Note: The subject must be provided a signed co of this document. |
| 1.2 | Demographics | Record the subject's year of bi1th, age, oender, race and ethnicit. |
| 1.3 | Medical Histoly and<br>Concomitant<br>Medications | Record the subject's medical histo1y and concomitant medic.ations. |
| 1.4 | Habitual Lenses | Record the subjects habitual lens type, parameters, lens care solution, wear modality, dmation of lens wear, and approximate rescrition date. |

| | Visit 1: Screenin | |
|---|---|---|
| Step | Procedure | Details |
| 1.5 | Eligibility after<br>Screening | AH responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |
| | | If subject is deemed to be ineligible after screening, proceed to Fina! Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms do not need to be completed as art o Fina! Evaluation. |

| | | Visit 1: Baseline |
|---|---|---|
| Step | Procedure | Details |
| 1.6 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual spectacle. Subjects must read the smallest line until at least 50% of the letters are read incon ectl. |
| 1.7 | Subjective Sphero-<br>cylindrical<br>Refraction | Complete subjective spherocylindrical refraction and record the resultant distance visual acuity (OD, OS, and OU) to the nearest letter. |
| 1.8 | Eye Dominancy | The investigator will detennine eye dominancy of the subject by first using the +1.00 blur test. If this fails to detennine dominancy, then the sighting test will be used. |
| 1.9 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If any of these slit lamp findings are grade 3 or higher, the subject may not continue at this time, but may return up to one additional time to detennine eligibility. If discontinued a final examination must be completed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline ma be instilled. |

| | | Visit 1: Baseline |
|---|---|---|
| Step | Procedure | Details |
| 1.10 | Eligibility after B ase line | AH responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. |
| | | If subject is deemed to be ineligible after baseline, proceed to Fina! Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms do not need to be com_leted_as_art_o Fjna! Evaluation. |

| | Visit 1: Treatment 1 Lens Fittin | |
|---|---|---|
| Step | Procedure | Details |
| 1.11 | Lens Selection | Assign the study lens based on the randomization scheme provided by the biostatistician. Select the contact lens power based on veltexed spherical equivalent from the refraction. |
| 1.12 | Lens Inse1tio11 | The Investigator or the subject inse1ts the study lenses. Record the time of lens inse1tio11. Check for lens damage under the slit lamp before proceeding with lens settling. Re lace damage delenses if a dicable. |
| 1.13 | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 1.14 | Subjective Best<br>Sphere Over<br>Refraction | Perfo1m subjective best sphere refraction over the study lenses (adopt the maximum plus to maximum visual acuity (MPMVA) a roach. |
| 1.15 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refractionis not plano. For each power modification, select the adjusted fitting lens power as appropriate and repeat steps 1.12 through 1.14. Up to two power modifications are allowed ere e. |

| | Visit I: Treatment I Lens Fittin | |
|---|---|---|
| Step | Procedure | Details |
| 1.16 | Subject Reported Ocular S m toms | Subjects will respond to a verbal open-ended s m toms uestionnaire. |
| 1.17 | Visual Acuity | Record the best conected Snellen distance visual acuity to the nearest letter (OD, OS and OU). Subjects must read the smallest line until at least 50% of the letters are read incon ectly. Visual acuity with the study contact lenses must be 20/30 or better OD and OS. |
| 1.18 | General Lens Fit<br>Assessment | Evaluate lens centration, movement on blink, a.ud push -up test for each eye. An unacceptable fit is deemed by one of the following criteria: Iimba! exposure at primalygaze or with extreme eye movement. edge lift. excessive movement in primaiy and up gaze. insufficient movement in all three of the following conditions: primaiy gaze, up gaze, and push-up test. |
| | | <b>Note:</b> if lens fit is unacceptable for either eye, the subject will be discontinued from the stud. |
| 1.19 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS. 2. The lens fit is acceptable OD and OS. 3. Investigator approval. If the Investigator does not approve the study lens, then the study is terminated for that subject. |

| Visit I : Treatment I Lens Fittin | | |
|---|---|---|
| Step | Procedure | Details |
| 1.20 | Lenses Wom in<br>Clinic | The lenses will be released for approximately two hours. 1. The subjects must wear both study lenses the entire time. 2. The lenses will be wom as daily wear only. 3. Rewetting drops are pennitted if needed. Note: In the event a lens is lost or damaged, it will be replaced immediately. A clinic-only-wear Patient Instruction Guide will be provided. |

Based on the randomization scheme, subjects are either in the photopic testing group or the mesopic testing group. Proceed to the coITect test:

| | | Visit I: Photo pic Testing |
|---|---|---|
| Step | Procedure | Details |
| 1.21 | Photopic Contrast<br>Sensitivity Testing<br>Without Glare | Contrast sensitivity testing will be perfo1med using the University of Georgia system OD and OS in the following order. The eye not being tested will be patched. The following spatial frequencies will be randomized: 1.6, 3.2, 8, 16 and 24 cpd. |
| | | Photopic contrast sensitivity without glare 1. Participant is seated in front of the optical device with their chin in the chin rest assembly and asked to patch OS. 2. To practice, the paiticipant is shown the 0.5 cycles per mm grating (which yields a threshold at 8 cycles per degree of visual angle). The procedure is demonstrated, and the paiticipant confinns that they can view the grating easil. |

| | | Visit 1: Photopic Testing |
|---|---|---|
| Step | Procedme | Details Details |
| | | <ol> <li>The pailicipant rests for a period of two minutes while the researcher replaces the 0.5 cycles per mm filter with the first spatial frequency grating dictated by the randomization scheme. Three ascending and three descending thresholds are obtained for the first spatial frequency dictated by the randomization scheme. EDC to record contrast sensitivity to 2 decimal places (range 0.01 - 10,000).</li> <li>The pailicipant rests for two minutes while the researcher changes the spatial frequency grating.</li> <li>The procedure is repeated until all 5 spatial frequencies have been tested, with two-minute breaks between trials. EDC to record contrast sensitivity to 2 decimal places (range 0.01 - 10,000). Area tmder the contrast sensitivity curve will be computed (range 5.00 - 20,000) and entered.</li> <li>The participant will then be given a 5-minute break and asked to change the patch to OD, in order to test OS.</li> <li>The procedure above will be repeated OS.</li> </ol> |
| 1.22 | Photopic Contrast<br>Sensitivity Testing<br>With Glai·e | Contrast sensitivity testing will be perfo1med using the University of Georgia system OD and OS in the following order. The eye not being tested will be patched. The following spatial frequencies will be randomized: 1.6, 3.2, 8, 16 and 24 cpd. |
| | | <ol> <li>The paiiicipant will be given a 5 minute break to change the patch back to OS while the researcher confinns alignment with the glare stimulus.</li> <li>The paiiicipailt will be instructed to keep eyes closed, and to position their chin in the chin rest assembl .</li> </ol> |

| Ctore | Duo oo daana | Visit 1: Photopic Testing |
|---|---|---|
| Step | Procedure | Details |
| | | 3. With the glare stimulus on, pailicipants will complete three ascending and three descending trials for the first spatial frequency dictated by the raildomization scheme for the glare condition. Note that the first spatial frequency tested in the glaire condition will likely be different from the first spatial frequency tested in the 110-gl are condition. EDC to record contrast sensitivity to 2 decimal places (range 0.01 - 10,000). 4. The pailicipant will be given a four minute break and will be instructed to keep eyes closed during the break. 5. The procedure is repeated until all 5 spatial frequencies have been tested, with four-minute breaks between trials. EDC to record contrast sensitivity to 2 decimal places (range 0.01 - 10,000). Area under the contrast sensitivity curve will be computed (range 5.00 - 20,000) and entered. 6. The pailicipant will then be given a 5-minute break and asked to change the patch to OD, in order to test OS. 7. The procedure above will be repeated |
| 1.23 | Lens Removal | OS. The wom study lenses will be removed and |
| 1.23 | Lons Removal | discarded. Proceed to the Final Evaluation. |

| | Visit 1: Mesopic Testing | |
|---|---|---|
| Step | Procedure | Details |
| 1.24 | Mesopic Contrast<br>Sensitivity Testing<br>Without Glare | Mesopic contrast sensitivity testing will be perfo1med using the University of Georgia system OD and OS in the following order. The eye not being tested will be patched. The following spatial frequencies will be randomized: 1.6, 3.2, 8, 16 and 24 cpd. |

| | Visit 1: Mesopic Testing | |
|---|---|---|
| Step | Procedme | Details |
| | | Mesopic contrast sensitivi ty without glare 1. Prior to seating the participant, the reseal cher confams that the wedge controlling the background luminance is dimmed to the appropriate position for mesopic testing. 2. Paiticipant is seated in front of the optical device with their chin in the chin rest assembly and asked to patch OS. 3. To practice, the participallt is shown the 0.5 cycles per mm grating (which wields a threshold at 8 cycles per |
| | | yields a threshold at 8 cycles per degree of visual angle). The procedure is demonstrated, and the palticipant confums that they can view the grating easily. 4. The pait icipant rests for a period of two minutes while the reseai cher replaces the 0.5 cycles per mm filter with the first spatial frequency grating dictated by the randomization scheme. Three ascending and three descending thresholds are obtained for the first spatial frequency dictated by the randomization scheme. EDC to record contrast sensitivity to 2 |
| | | decimal places (range 0.01 - 10,000). 5. The paiticipant rests for two minutes while the reseai cher changes the spatial frequency grating. 6. The procedure is repeated until all 5 spatial frequencies have been tested, with two-minute breaks between trials EDC to record contrast sensitivity to 2 decimal places (range 0.01 - 10,000). Area under the contrast sensitivity cmve will be computed (range 5.00 - |
| | | 20,000) and entered. 7. The participant will then be given a 5-minute break and asked to change the atch to OD, in order to test OS. |

| | Visit 1: Mesopic Testing | |
|---|---|---|
| Step | Procedure | Details |
| | | The procedure above will be repeated OS. |
| 1.25 | Mesopic Contrast<br>Sensitivity Testing<br>With Glai-e | Mesopic contrast sensitivity testing will be perfol med using the University of Georgia system OD and OS in the following order. The eye not being tested will be patched. The following spatial frequencies will be randomized: 1.6, 3.2, 8, 16 and 24 cpd. Mesopic contrast sensitivity with glare 1. Prior to seating the pariicip ant, the researcher confirms that the wedge controlling the background luminance is dimmed to the appropriate position for mesopic testing. 2. The pariicipant will be given a 5 minute break to change the patch back to OS while the researcher confinns alignment with the glare stimulus. 3. The pariicipant will be instructed to keep eyes closed, and to position their chin in the chin restassembly. 4. With the glare stimulus on, pariicipants will complete three ascending and three descending trials for the first spatial frequency dictated by the randomization scheme for the glare condition. Note that the first spatial frequency tested in the glare condition will likely be different from the first spatial frequency tested in the no-glare condition. EDC to record contrast sensitivity to 2 decimal places (range 0.01 - 10,000). 5. The pariicipant will be given a four minute break and will be instructed to keep eyes closed during the break. 6. The procedure is repeated until all 5 spatial frequencies have been tested, with four-minute breaks between trials. EDC to record contrast |
| | | sensitivity to 2 decimal laces range |

| | Visit 1: Mesopic Testing | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>0.01 - 10,000). Area under the contrast sensitivity curve will be computed (range 5.00 - 20,000) and entered.</li> <li>7. The participant will then be given a 5-minute break and asked to change the patch to OD, in order to test OS.</li> <li>8. The procedure above will be repeated OS.</li> </ul> |
| 1.26 | Lens Removal | The wom study lenses will be removed and discarded. Proceed to the Final Evaluation. |

### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is tenninated from the study.

| | Final Evaluation | |
|---|---|---|
| Ste | Procedure | Details |
| F.1 | Final Exam Fo1m | fudic ate if the subject completed the study successfully. If subject discontinued from the stud indicate the reason. |
| F.2 | Exit Slit Lamp<br>Bioinicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. This step is not necessaly if the subject was exited due to screen failure. |
| F.3 | Exit Visual Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual con ection in place. Subjects must read the smallest line until at least 50% of the letters are read inconectl. |

#### 7.3. UnscheduledVisits

If , during the investigation, a subject requires an unscheduled visit to the clinical site, the following info1mation will be collected, as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test aiticle dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report fo1ms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that ai-e ongo ing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If fmther treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health cai e provide r.

The following info1m ation will be collected dming an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Ste | Procedme | Details |
| U.I | Reason for unscheduled visit | Indicate if the <u>only</u> reason for the visit is that the subject requires additional test aiticles. If the reason is other than resupply of previously dispensed lenses, specify the reason for the visit. |
| U.2 | Chief Complaints (if a lic.able | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.3 | Adverse Events and Concomitant Medications Review if a licable | Review any changes to the subject's medica! histoly or concomitant medications from the previous study visit. Record any changes, and an adverse events. |
| U.4 | Entrance VA (if a licable | Record the entrance distance visual acuity OD, OS, and OU to the nearest letter. |
| U.5 | Subjective Sphero-<br>cylindrical<br>Refraction (if<br>applicable) | Perfolm bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best conected <u>distance</u> visual acuity to the nearest letter OD OS, and O |

| | Unscheduled Visit | |
|---|---|---|
| Ste | Procedure | Details |
| U.6 | Slit Lamp<br>Biomicroscopy (if<br>applic.able) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.7 | Dispensing(if applicable) | If the subject requires additional lenses to complete the wear period and is eligible to do so, previde additional lenses per the dispensing instructions given in the detailed stud rocedures. |
| U.8 | Exit Visual Acuity if a licable | Record the subject's exit distance visual acm OD, OS, and O to the nearest letter. |

NOTE: If the only reason for the unscheduled visit is that the subject requires additional test aiticles, only the dispensing infonnation needs to be recorded.

### 7.4. Laboratory Procedures

None

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

### 8.1. Completion Criteria

Subjects are considered to bave completed the study if they:

- provided info1med consent.
- they ai e eligible.
- Complete d a ll sc hedu led tests

#### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the shldy for any of the following reasons:

- Subject withdrawal of consent.
- Subject not compliant to protocol (e.g., subject does not complete all scheduled tests).
- Subject develops significant or serious adverse events necessitating discontinuation of study lens wear.
- Subjects who have experienced a Comeal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject not successfully released with lenses due to lack of efficacy and safety including poor vision, poor comfolt or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) from the subject and discard them, unless otherwise stated in section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

Additional subjects will be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: any ocular medications. Concomitant therapies that are disallowed include: see section 9.1.

#### 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film.

A summary of disallowed systemic medications is shown in Table 4. Subjects with a history of taking these medications will be allowed to enroll only if:

- The medications have been taken on a continual, routine basis for at least 6 months, and
- The subject has demonstrated successful contact lens wear during this time.

Or:

• The subject was taking the medication on a temporary basis and ceased taking that medication at least 2 weeks prior to signing the informed consent (this is considered sufficient time for the medication to have left the body prior to enrollment).

Subjects with a history of taking medications listed in Table 4 on a long-term, routine basis for less than 6 months will not be allowed to participate in the study.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Estrogens (not including contrnceptive medication) | Menopause, osteoporosis, vaginitis | Vagifem, Estrace, Climara, Vivelle-Dot, Premarin, Minivelle, etc. |
| Anticholinergics | IITitable bowel syndrome,<br>Parkinson's disease, peptic ulcer,<br>cystitis, nasal congestion, cold<br>symptoms, overactive bladder,<br>COPD | Hyosyne, Levsin, Symax Fastab,<br>Symax SL, Homax SL, Cogentin, |
| Beta-blockers | Hypertension, angina, heait attack, migraine, atrial fibrillation, adrenal cancer, essential tumor, glaucoma | Toprol XL, Lopressor, Tenonnin, Propranolol, Timoptic, Trandate, Inderal LA, etc. |
| Psychotropics | Antipsychotic (schizophrenia, mania), antidepression, antiobsessive, antianxiety, mood stabilizer, stimulants (ADHD) | Zoloft, Celexa, Prozac, Lexapro,<br>Effexor, Cymbalta, Ativan,<br>Xanax, Desyrel, Wellbutrin, etc. |
| Vitamin A analogs | Cystic acne | Isotretinoin |

Examples of disallowed systemic antihistamines are given in Table 5. Subjects with a histoly of taking systemic antihistamines will be allowed to emoll only if:

- They have taken antihistamines continuously for at least 2 weeks, and
- They have demonstrated successful weai while taking the medication

Or:

• They stopped taking the medication for at least 2 weeks prior to emollment.

Table 5: Disallowed systemic antihistamines

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Antihistamines | Allergic rhinitis, sedation, hives, | |
| | allergic conjm1ctivitis, skin allergy, | |
| | itching, motion sickness | Zyitec, Astepro, Astelin, Optivar, |
| | | Allegra, Benadiyl, etc. |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovely of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.


If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigatormust notify and provide the rationale to the Sponsor and as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations that contradict the infolmation contained in the Infolmed Consen/tAssent folms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They ai e often logistical in nature.

Protocol waivers are prohibited.

Table 6 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 6: Examples of major and minor protocol deviations

| <b>Deviation category</b> | Major deviation | Minor deviation |
|---|---|---|
| Incomplete tests | Subject does not complete all scheduled psychophysical tests. | |

In the case of a major protocol deviation, the decision of whether or not the subject will be excluded from the Per-Protocol analysis population will be made at the time of coholt review.

#### 11. STUDY TERMINATION

The occunence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be mled out, may result in stopping fmther dispensing of test alticle. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any fmther subjects are enrolled.

The Sponsor will detennine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if infolmation indicates the study's results are compromised.

JJVC reserves the right to telminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to telminate the study if an unreasonable risk is detelmined. The study can be telminated by the Principal Investigator at the individua! clinical site due to

specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).

- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also apply and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** - An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated."

**Note**: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

**Note**: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) - An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Foetal distress, foetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** - are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** - are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** - An ADE is an "adverse event related to the use of an investigational medical device."

NOTE 1: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

NOTE 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.<sup>1</sup>

**Unanticipated Adverse Device Effect (UADE)** - A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related, unlikely related, possibly related, or related see definition in section 13.2.1).

- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in section 13.2.2).
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

### 13.2.1. Causality Assessment

**Causality Assessment** - A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

### 13.2.2. Severity Assessment

**Severity Assessment** - A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be

recorded as medical history. However, if the condition deteriorates at any time during the study, it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review formust be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as

intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

## 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

### 13.4.1. Reporting Adverse Events to Sponsor

#### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.

- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according to the written guidelines, including reporting timelines.

## 13.5. Event of Special Interest

None.

#### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

## 14.2. Sample Size Justification

The plan is to enroll approximately 44 subjects with approximately 40 subjects to compete the study. Given that no historical data is available for the primary and secondary endpoints using the same glare system, the sample size was not determined based on any empirical sample size calculation. Targeting 40 subjects to complete the study (20 subjects for each condition arm) is considered appropriate to assess descriptive summaries of the primary and secondary endpoints. The data collected for this study may be used to design future clinical trials.

## 14.3. Analysis Populations

The following analysis populations will be defined and used in the analysis and presentation of the data.

#### All Enrolled:

All Enrolled Population includes all subjects with recorded data in the electronic Case Report Form (eCRF) database.

#### **Safety Population:**

All subjects who are administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded. Subjects will be analyzed as per treatment received.

#### **Per-Protocol Population:**

All subjects who successfully complete all visits and do not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock.

Justification for the exclusion of subjects with protocol deviations from the per-protocol population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol. At least one observation should be recorded. Subjects will be analyzed as per randomized treatment.

## 14.4. Level of Statistical Significance

No primary or secondary hypothesis will be tested. Each exploratory hypothesis will be tested at the 2-sided Type I error rate of 0.05.

### 14.5. Primary Analysis

No primary hypothesis will be tested. The primary endpoint will be summarized descriptively, as discussed in 14.1.

### 14.6. Secondary Analyses

No secondary hypothesis will be tested. The secondary endpoint will be summarized descriptively, as discussed in 14.1.

## 14.7. Other Exploratory Analysis

Exploratory analyses of the primary and secondary endpoints will be conducted using the ITT population. With a broadband glare source, the AUC of the photopic and mesopic contrast sensitivity function will be analyzed separately using a linear mixed effects model. Lens type, dominant eye, and the interaction of lens type by dominant eye will be included in the model as fixed effects adjusting for age and gender. The covariance of residuals of within-subject repeated measurements (R-side) will be modeled using Unstructured (UN) covariance structure. If the model does not converge, then a compound Symmetry (CS) covariance structure will be considered. The Kenward and Roger method will be used for the denominator degrees of freedom.<sup>8</sup>

## Hypothesis Testing

The null and alternative hypotheses for testing superiority of the Test Lens compared to the Control lens from the previously described model are presented below:

$$H_0 \mu_T - \mu_C > 0$$
  
 $H_A \mu_T - \mu_C > 0$ 

Where,  $\mu_T$  and  $\mu_C$  represent the mean AUC of photopic or mesopic contrast sensitivity function with a glare source for the Test lens and the Control lens, respectively. Statistical superiority will be declared if the lower bound of the 2-sided 95% confidence interval of the mean difference (Test - Control) is larger than 0. A model-based point estimate of the mean difference being 0.06 log or more (2'0.06 log) will be considered clinically meaningful.

If the proposed mixed effect model fails to converge, the hypothesis will be tested using a paired sample *t*-test or equivalent non-parametric method.

Other study endpoints and observations will be summarized descriptively. Further exploratory and/or post-hoc analyses may be conducted at the discretion of the study responsible clinician.

### 14.8. Interim Analysis

Not applicable.

## 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

## 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The vision assessments (photopic and mesopic contrast sensitivity with and without glare) will be collected using the previously validated optical device described above. The data from the device will be recorded on a paper case report form (CRF) stored at the study site. Paper forms will be used to record the raw values that are used to compute the final sensitivity values, which are then entered into electronic case report forms (eCRFs) using the Bioclinica EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of

the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2020.<sup>1</sup>

### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by

the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 16.4. Data Monitoring Committee (DMC)

Not applicable

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.

• Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study, and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Subjects will only be enrolled if the subject is fully able to understand the risks, benefits, and potential adverse events of the study and provide their consent voluntarily.

### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, according to ISO 14155:2020, and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>2</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>2</sup> and ISO 14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

## 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.
Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ISO 14155:2020,<sup>1</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ISO 14155:2020<sup>1</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

This is a single site study. The participating institution and Principal Investigators for this study agree that, should the study results be published, the first publication of the results of this study shall be made in conjunction with the presentation of a joint publication of the study results with the investigators contributing data, analyses and comments.

#### 22. REFERENCES

- 1. ISO 14155:2020: Clinical investigation of medical devices for human subjects Good clinical practice, Available at: https://www.iso.org/standard/71690.html
- 2. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects, Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 3. United States (US) Code of Federal Regulations (CFR). Available at https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 4. Buch J. The Effects of Contact Lenses With HEV-Blocker on Visual FunctionAugust 21, 2019.
- 5. Buch J. The Effects of Contact Lenses With UV/HEV-Blocker on Visual FunctionJune 22, 2021.
- 6. Kojima T HA, Hara S, et al. Quantitative evaluation of night vision and correlation of refractive and topographical parameters with glare after orthokeratology. *Graefe's Archive for Clinical and Experimental Ophthalmology*. 2011;249(10):1519-1526.
- 7. SAS/STAT® 14.3 User's Guide. Cary, NC: SAS Institute Inc; 2016.

- 8. Kenward MG, Roger JH. An Improved Approximation to the Precision of Fixed Effects from Restricted Maximum Likelihood. *Computational Statistics and Data Analysis*. 2009(53):2583-2595.
- 9. Health Information Portability and Accountability Act (HIPAA), Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)

Not Applicable for this study.

### APPENDIX B: PATIENT INSTRUCTION GUIDE

Not Applicable for this study.

APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

#### **PACKAGE INSERT & FITTING INSTRUCTION GUIDE**



#### **ACUVUE® OASYS MAX 1-Day Contact Lenses**

#### **ACUVUE® OASYS MAX 1-Day MULTIFOCAL Contact Lenses**

senofilcon A Soft (hydrophilic) Contact Lenses for Daily Disposable Wear

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at <a href="https://www.acuvue.com">www.acuvue.com</a>.



CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

### SYMBOLS KEY

The foll owing symbols may appear on the labelor carton:

| SYMBOL | DESCRIPTION |
|---|---|
| &(D) | Caution, Consult Inst ructio ns for Use |
| d | Date of Manufacture |
| • • | Manufacturer |
| | Use-By Date (expiration date) |
| | Batch Code |
| 'ЮLII11 | Sterilized Using Steam Heat |
| | Indicates a Single Sterile Barrier System |
| DIA | Diameter |
| ВС | Base Curve |
| D | Diopter (lens power) |
| <b>CE:</b> 2191 | CE Mark and lde nti fication number of Notified Body |
| UV BLOCKIN G | UV Blocking |
| e) | Fee Paid for Waste Management |
| <u>l</u> <u>Oriy</u> | CAUTION: US Federal law restricts this device to sale by or on the order of a licensed practitioner |
| | Lens Orientation Correct |
| X | Lens Orientation Inco rrect<br>(Lens Inside Out) |
| EC j R EP | Authorized Representative in the European Community |
| | Contains Hazardous Substances |
| R | Do Not Re -Use (Single<br>Use) |
| | Do Not Use if Package is Damaged |
| | Medical Device Symbol |
| • • | Package Opening Icon (Blister) |
| G | Package Opening Icon (Carton) |
| L | "Low" near ADD |
| M | "Medium" near ADD |
| Н | "High" near ADD |
| MAXADD | Near ADD |

## **Clinical Study Protocol**

CR-6501, v 4.0

| LOW | "Low" near ADD |
|-----|-------------------|
| MID | "Medium" near ADD |
| HGH | "High" near ADD |

Visit www.acuvue.com/guides for additional information about symbols.

#### **DESCRIPTION**

ACUVUE® OASYS MAX 1-Day Contact Lenses are soft (hydrophilic) contact lenses available as spherical and multifocal lenses.

These lenses are made of a silicone hydrogel material (senofilcon A) containing an internal wetting agent and are tinted using Reactive Blue Dye #247 to make lenses more visible for handling.

A benzotriazole ultraviolet (UV) absorbing monomer is used to block UV radiation (280 nm - 380 nm) in combination with a novel fused tricyclic chromophore that also blocks UV radiation and partially filters high energy visible radiation (HEV)\* in the range of 380 nm to 450 nm. The light transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and 10% in the UVA range of 315 nm to 380 nm. The thinnest lenses transmit � 45% of the radiation in the range from 380 nm to 450 nm. Please see HEV filtering NOTE in the ACTIONS section below.

#### **Lens Properties:**

The physical/optical properties of the lens are:

Specific Gravity (calculated): 0.98 - 1.12
 Refractive Index: 1.42
 Visible Light Transmittance: ;?78%
 HEV Light Transmittance\*: 45%
 Surface Character: Hydrophilic

• Water Content: 38%

Oxygen Permeability (Dk):

VALUE METHOD

103 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, edge

(ml  $O_2$ /mL x mm Hg) @ 35°C corrected)

#### **Lens Parameter Ranges:**

Diameter (DIA): 12.0 mm to 15.0 mm

Center Thickness: varies with power

Base Curve (BC): 7.85 mm to 10.00 mm
 Spherical Power (D): -20.00D to +20.00D
 Multifocal ADD Power: +0.25D to +4.00D

Each lens is supplied in a foil-sealed plastic package containing borate buffered saline solution with methyl ether cellulose.

#### **AVAILABLE LENS PARAMETERS**

The ACUVUE® OASYS MAX 1-Day Contact Lenses (senofilcon A) are hemispherical shells of the following dimensions:

Diameter (DIA): 14.3 mm

**Center Thickness:** 0.085 mm to 0.221 mm (varies with power)

Base Curve (BC): 8.5 mm, 9.0 mm

**Powers (D):** -12.00D to +8.00D

The ACUVUE® OASYS MAX 1-Day MULTIFOCAL Contact Lenses (senofilcon A) are hemispherical shells of the following dimensions:

Diameter (DIA): 14.3 mm

**Center Thickness:** 0.070 mm to 0.191 mm (varies with power)

Base Curve (BC): 8.4 mm

**Powers (D):** -9.00D to +6.00D

**ADD Powers (D):** +1.25D (LOW), +1.75D (MID), +2.50D (HGH)

#### TRANSMITTANCE CURVE

ACUVUE® OASYS MAX 1-Day Contact Lenses (senofilcon A) vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



<sup>1</sup> Le r man, S., Rad ia nt Energy and the Eye, MacMillan, Ne w York, 1980, p. 58, figure 2-21 <sup>2</sup>Waxler, M. Hitchins, V.M., Optica l Radiation and Vis ua l Health, CRC Press, Boca Raton, Flor ida, 1986, p. 19, figure S

#### **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays on the retina.

These lenses contain UV and HEV\* light absorbing monomers to help protect against transmission of harmful UV radiation to the cornea and into the eye and reduce transmittance of HEV\* light. The light transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 315 nm to 380 nm for the entire power range. The thinnest lenses transmit \$ 45% of the radiation across the high energy visible\* light wavelength in the range from 380 nm to 450 nm. The visible light transmittance in the range from 380 nm to 780 nm is greater than or equal to 78% depending on the lensthickness.

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. You should continue to use UV absorbing eyewear as directed.

NOTE: long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography,

<sup>&</sup>lt;sup>3</sup>The data wasobtained from measurements taken through the centra I 6 mm portion for the thinne st sing le vision le ns (-0.500 lens, 0.085mm center thickness).

## **Clinical Study Protocol**


cloud cover) and personal factors (extent and nature of outdoor activities). UV Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

\*NOTE: Filtering of HEV light by contact lenses has not been demonstrated to confer any health benefit to the user, including but not limited to retinal protection, protection from cataract progression, reduced eye strain, improved contrast, improved acuity, reduced glare, improved low light vision, or improved circadian rhythm/sleep cycle. The Eye Care Professional should be consulted for more information.

#### INDICATIONS (USES)

ACUVUE® OASYS MAX 1-Day Contact Lenses (senofilcon A) are indicated for daily disposable wear for the correction of vision in people with non-diseased eyes who are nearsighted (myopic) or farsighted (hyperopic) and may have 1.00D or less of astigmatism that does not interfere with visual acuity.

ACUVUE® OASYS MAX 1-Day MULTIFOCAL Contact Lenses (senofilcon A) are indicated for daily disposable wear for the correction of vision in people with non-diseased eyes who are presbyopic and may be nearsighted (myopic) or farsighted (hyperopic) and may have 0.75D or less of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for daily disposable wear. Therefore, no cleaning or disinfection is required. Lenses should be discarded upon removal.

#### **CONTRAINDICATIONS (REASONS NOT TO USE)**

DO NOT USE these lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye
- Any eye disease, injury or abnormality that affects the cornea, conjunctiva, or eyelids
- Severe insufficiency of lacrimal secretion (dry eye)
- Corneal hypoesthesia (reduced corneal sensitivity)
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses
- Ocular irritation due to allergic reactions which may be caused by use of contact lens solutions (i.e. rewetting drops) that contain chemicals or preservatives (such as mercury or Thimerosal, etc.) to which some people may develop an allergic response
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses
- Any active corneal infection (bacterial, fungal, protozoal, or viral)
- If eyes become red or irritated

#### **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION. IF THE PATIENT EXPERIENCES:

- Eye Discomfort,
- Excessive Tearing,
- Vision Changes,
- Loss of Vision,
- Eye Redness, or
- Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES, AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

- Patients should be instructed not to wear their lenses while sleeping. Clinical studies have shown that the risk of serious adverse reactions is increased when lenses are worn overnight, and that the risk of ulcerative keratitis is greater for extended wear contact lens users than for daily wear users.<sup>4</sup>
- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye.
   Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.
- The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

<sup>4</sup>New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

#### **Specific Instructions for Use and Warnings:**

Water Activity

Instruction for Use

Do not expose contact lenses to water while wearing them.

#### **WARNING:**

Water can harbor microorganisms that can lead to severe infection, vision loss, or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

#### **PRECAUTIONS**

#### **Special Precautions for Eye Care Professionals:**

- Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.
  - The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.
- Patients who wear these lenses to correct presbyopia using monovision or multifocal correction may not achieve the best corrected visual acuity for either far or near vision.
   Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes unless
  otherwise indicated. The lenses absorb this dye and become discolored. Whenever
  fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is
  recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove lenses immediately if the eyes become red or irritated.

Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions:

#### **Handling Precautions:**

- Before leaving the Eye Care Professional's office, the patient should be able to promptly
  remove lenses or should have someone else available who can remove the lenses for him or
  her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash, rinse, and dry hands before handling lenses. It is best to put on lenses before putting on makeup.
- DO NOT touch contact lenses with fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the "Patient Instruction Guide" for ACUVUE® OASYS MAX 1-Day Contact Lenses and those prescribed by the Eye Care Professional.
- Always handle lenses carefully and avoid dropping them.

• Never use tweezers or other tools to remove lenses from the lens container. Slide the lens up the side of the bowl until it is free of the container.

#### **Lens Wearing Precautions:**

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for a Sticking (Non-Moving) Lens". The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.
- The patient should be advised to never allow anyone else to wear their lenses. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hair spray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.
- Ask the Eye Care Professional about wearing lenses during sporting activities.
- The patient should be advised to never rinse the lenses in water from the tap. Tap water contains many impurities that can contaminate or damage the lenses and may lead to eye infection or injury.

#### **Lens Care Precautions:**

• The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

#### Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed. Depending on the severity, this could include the use of lubricating drops that are indicated for use with soft contact lenses or the temporary discontinuance of contact lens wear while such medication is being used.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- Do not change lens type (e.g. brand name, etc.) or parameters (e.g. diameter, base curve, lens power, etc.) without consulting the Eye Care Professional.
- Instruct patients to always confirm the lens parameters printed on the multi-pack and on the individual lens package match their prescription. If there is a mismatch the patient should not use the product.

 As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

#### Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

#### **ADVERSE REACTIONS**

The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may burn, sting and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis; some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions or redness of the eye.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry
  eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to

seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.

#### **GENERAL FITTING GUIDELINES**

#### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- Motivation to wear lenses
- Ability to follow instructions regarding lens wear care
- General health
- Ability to adequately handle and care for the lenses
- Ability to understand the risk and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses.

#### B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the appropriate lens fitting instruction outlined below.

#### C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if necessary.

#### D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, corneal curvature measurements should be performed to establish the patient's baseline ocular status.

For the Spherical or Multifocal ACUVUE® OASYS MAX 1-Day Contact Lenses, the initial lens should be selected from the currently available base curves.

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

#### 1. Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

#### 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink, and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

#### 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

#### E. Final Lens Power

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

| Example 1: | | |
|------------------|----------------------------|--------|
| Diagnostic lens: | | -2.00D |
| | Spherical over-refraction: | -0.25D |
| | Final lens power: | -2.25D |

| Example 2: |
|------------|

| Diagnostic lens: | | -2.00D |
|------------------|----------------------------|--------|
| | Spherical over-refraction: | +0.25D |
| | Final lens power: | -1.75D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see dispensing and follow up information in **PATIENT MANAGEMENT**).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download from <a href="https://www.acuvue.com">www.acuvue.com</a>.

#### **MULTIFOCAL FITTING GUIDELINES**

#### A. Presbyopic Needs Assessment & Patient Education

Multifocal contact lenses may produce compromise to vision under certain circumstances and the patient should understand that they might not find their vision acceptable in specific situations (i.e., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments. Occupational and environmental visual demands should be considered. If the patient requires critical visual acuity and stereopsis, it should be determined by trial whether this patient can function adequately with the ACUVUE® OASYS MAX 1-Day Multifocal Contact Lenses. Wear may not be optimal for such activities as:

- 1. Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- 2. Driving automobiles (e.g., driving at night). Patients who cannot pass their state driver's license requirements with these lenses should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

These lenses are not recommended for patients who have -1.00D or greater of refractive cylinder as this level of uncorrected cylinder may lead to additional visual compromise.

These lenses are available in the following ADD powers:

- Lens "LOW" ="low" near ADD lens (Max +1.25 ADD)
- Lens "MID" = "medium" near ADD lens (Max +1.75 ADD)
- Lens "HGH" = "high" near ADD lens (Max +2.50 ADD)

#### **B.** Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is ;? ±4.00D. Determine the spherical equivalent distance prescription for a multifocal patient. Determine the eye dominance using one of the methods below:

<u>Method 1:</u> Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

<u>Method 2 (preferred):</u> Determine which eye will accept the added power with the least reduction in vision while both eyes are open. Place a hand-held trial lens equal to +1.00D in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the +1.00D lens over the right or left eye, which is the non-dominant eye.

#### C. Select the Initial Trial Lens

- 1. For each eye, select the trial lens distance power that is closest to the patient's distance spherical equivalent. Remember to compensate for vertex distance if the refraction is ;? ±4.00D.
- Select the near power of the lens based on the patients ADD range as follows:
  - ADD: +0.75 to +1.25 use a "LOW" near ADD lens on each eye
  - ADD: +1.50 to +1.75 use a "MID" near ADD lens on each eye
  - ADD: +2.00 to +2.50 use a "MID" near ADD on the dominant eye and a "HGH" near ADD lens on the non-dominant eye
- 3. Allow the lenses to settle for a minimum 10 minutes.
- 4. Assess distance and near vision binocularly and monocularly.
- Demonstrate the vision under various lighting conditions (normal and decreased illumination) and at distance, intermediate and near.
- 6. Make adjustments in power as necessary based on the distance over-refraction. The use of hand held trial lenses is recommended. Check the impact on distance and near vision.
- 7. If vision is still unacceptable, make adjustments in power as necessary (see "Multifocal Troubleshooting" below). If distance and near vision are acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).

#### D. Multifocal Troubleshooting

#### **Unacceptable Near Vision:**

If it has been determined that no change is required based on the over-refraction then add +0.25 D to the spherical power of the non-dominant eye.

#### **Unacceptable Distance Vision:**

If it has been determined that no change is required based on the over-refraction then make the changes as listed below:

- If the patient is wearing two "LOW" ADD lenses, change the dominant eye to an ACUVUE® OASYS MAX 1-Day Contact Lens sphere lens with a power equal to the spherical equivalent distance prescription.
- If the patient is wearing two "MID" ADD lenses, change the ADD power in the dominant eye to the "LOW" ADD power.

• If the patient is wearing a "MID" ADD lens in the dominant eye and a "HGH" ADD lens in the non-dominant eye, change the non-dominant eye to a "MID" ADD lens and add +0.25D to the distance power.

Once the changes have been made for the troubleshooting repeat steps 3-6 in section C above ("Select the Initial Trial Lens") to assess if the vision is acceptable.

#### E. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download from <a href="https://www.acuvue.com">www.acuvue.com</a>.

#### MONOVISION FITTING GUIDELINES

#### A. Patient Selection

#### **Monovision Needs Assessment**

For a good prognosis the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient with significant amounts of uncorrected astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

(1) visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and

(2) driving automobiles (e.g., driving at night). Patients who cannot pass their state driver's license requirements with monovision correction should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

#### **Patient Education**

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised. During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision, and straight ahead and upward gaze that monovision contact lenses provide.

#### **B.** Eye Selection

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

#### 1. Ocular Preference Determination Methods

Method 1: Determine which eye is the "sighting eye." Have the patient point to an object at

the far end of the room. Cover one eye. If the patient is still pointing directly at

the object, the eye being used is the dominant (sighting) eye.

Method 2: Determine which eye will accept the added power with the least reduction in

vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near

ADD lens over the right or left eye

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### 2. Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### 3. Visual Demands Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example:

A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

#### **C. Special Fitting Characteristics**

#### 1. Unilateral Vision Correction Requirement

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens whereas a bilateral myope would require corrective lenses on both eyes.

#### Example:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the "General Fitting Guidelines" for base curve selection described in this guide.

Case history and standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to news print and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches and a feeling of slight imbalance. You should explain the adaptation symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

#### S. Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Having supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet their state driver's license requirements with a monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Monovision fitting success can be improved with the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.

■ Emphasize the benefits of clear near vision and straight-ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download from <a href="https://www.acuvue.com">www.acuvue.com</a>.

#### **PATIENT MANAGEMENT**

- Follow the accepted standard of care in fitting and following up with your patient.
- Schedule the appropriate follow-up examination.
- Preferably, at the follow-up visits, lenses should have been worn for at least six hours.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses, which
  can be found at <a href="www.acuvue.com">www.acuvue.com</a>. REVIEW THESE INSTRUCTIONS WITH THE PATIENT SOTHAT
  HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT
  SCHEDULE (DAILY DISPOSABLE).

#### WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to over wear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

The maximum suggested wearing time for these lenses is:

| Day | Hours |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

#### REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

#### **LENS CARE DIRECTIONS**

When lenses are dispensed, the Eye Care Professional should provide the patient with appropriate and adequate warnings and instructions for daily disposable lens wear.

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with disposable lenses. Patients should always dispose of lenses when they are removed and have spare lenses or spectacles available.

#### **Basic Instructions:**

- Always wash, rinse, and dry hands before handling contact lenses.
- Do not use saliva or anything other than the recommended solutions for lubricating or rewetting lenses. Do not put lenses in the mouth.
- Eye Care Professionals may recommend a lubricating/rewetting solution which can be used to wet (lubricate) lenses while they are being worn to make them more comfortable.

#### Care for a Sticking (Non-Moving) Lens

During removal, if the lens sticks to the eye, the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should immediately consult the Eye Care Professional.

#### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

#### **REPORTING OF ADVERSE REACTIONS**

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with the lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA

Tel: 1-800-843-2020 www.acuvue.com

Revision Date: 02/2022

Revision Number: AO-01-22-03

IMPORTANT: Please read carefully and keep this Information fIN' future use.

This Package Insert and Frtting Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The EyeCare Professional should provide the patient wittl the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for **download** at www.acuvu.ecom.



ACUWE OASYS• Brand Contact lenses 1-Day witil HydraLuxeM Technology

ACUWE OASYS• Brand Contactlenses1-Day with Hydraluxe" Teclinology for ASTIGMATISM

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted withUV Blocker for Daily Disposable Wear

rii':n.i:7 CAUTION:U.S. Federallawrestricts this device to sale by or on the order of a licensed practitioner

## SYMBOLS KEY

The following symbols may appear on the label or carton:

| SYMBOL | DEFINITION |
|---|---|
| lliJ | Consult Instructions for Use |
| | Manufactured by or in |
| d | Date of Manufacture |
| | Use By Date (expiration date) |
| ILOTI | Batch Code |
| STERILE 1 | Sterile Using Steam or Dry Heat |
| R | Single-Use |
| DIA | Diameter |
| ВС | Base Curve |
| D | Diopter (lens power) |
| CYL | Cylinder |
| AXIS | Axis |
| <b>CE</b><br>0086 | Quality System Certification Symbol |
| I!)<br>∪∨ Blockin9 | UV-Blocking |
| (e) | Fee Paid for Waste Management |
| il <b>Jt</b> only l | CAUTION: U.S. Federa! law restricts this device to sale by or on the order of a licensed practitioner |
| 'lW <b>e</b> | Lens Orientation Correct |
| 'qD7<br>X X | Lens Orientation Incorrect (Lens Inside Out) |

### DESCRIPTION

ACUVUE OASYS® Brand Contact Lenses 1-Day and ACUVUE OASYS Brand Contact Lenses 1-Day for ASTIGMATING are soft (hydrophilic) contact lenses made with HydraluxerM TechnologyThey are available as spherical or toric lensesrespective.ly

These lenses are made of a siliconehydrogel material containing an interna! wetting agent, visibility tint, and UV absorbingmonomer and are tinted blue using Reactive Blue Dye #4 to make the lensesmore visible for handling.

A benzotriazole UV absorbing monomer is used to block UV radiation. The transmittance characteristics for these lensesare lessthan 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

#### **lens Properties:**

#### The physical/optical properties of the lens are:

| • | Specific | Gravity | (calculated) | ): 0.98 | - 1.12 |
|---|----------|---------|--------------|---------|--------|
|---|----------|---------|--------------|---------|--------|

RefractiveIndex: 1.42

85% minimum Light Transmission:

Surface Character: Hydrophilic

Water Content: 38%

Oxygen Permeability:

| VALUE | METHOD |
|-------|--------|
|-------|--------|

122 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, non-(mi O/ mi x mm Hg) at 35°C edge corrected) 103 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, edge corrected) (mi O/ mi x mm Hg) at 35°C

#### Lens Parameters:

Base Curve Range:

Diameter Range: 12.0 mm to 15.0 mm Center Thickness: varies with power 7.85 mm to 10.00 mm

-20.00D to +20.00D Spherical Power Range:

Cylinder Power Range: -0.25D to -10.00D

2.5° to 180° Axis Range:

### AVAILABLE LENS PARAMETERS

ACUVUE OASYS® Brand 1-Day with Hydraluxe<sub>TM</sub> Technology are hemispherical shells of the following dimensions:

**Diameter:** 14.3 mm

**Center Thickness:** 0.085 mm to 0.221 mm (varies with power)

Base Curve: 8.5 mm, 9.0 mm

**Powers:** -0.50D to -6.00D (in 0.25D increments)

-6.50D to -12.00D (in0.50D increments) +0.50D to +6.00D (in 0.25D increments) +6.50D to +8.00D (in0.50D increments)

ACUVUE OASYS® Brand 1-Day with Hydraluxe<sub>TM</sub> Technology for ASTIGMATISM are hemitoric shells of the following dimensions:

**Diameter:** 14.3 mm

**Center Thickness:** 0.075 mm to 0.172 mm (varies with power)

Base Curve: 8.5 mm

**Powers:** +0.00D to -6.00D (in 0.25D increments)

Cylinders: -0.75D, -1.25D, -1.75D, -2.25D\*

Axis: 10° to 180° in 10° increments

\*-2.25Dcylinder is availble in 10°, 20°, 70°, 80°, 90°, 100°, 110°,

160°, 170°, 180° axes only.

+ 0.25D to +4.00D (in 0.25D increments)

-6.50D to -9.00D (in 0.50D increments)

Cylinders: -0.75D, -1.25D, -1.75D

Axis: 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

### TRANSMITTANCE CURVES

ACUVUE OASYS® 1- Day with Hydraluxe™ Technology (senofilcon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



ACUVŒ 0ASY®

1-Daywith
Hydraluxe™
Technology
(senofilconA)\*

24 YR. OLD HUMAN
CORNEA¹

25 YR. OLD HUMAN CRYSTALLINE LEN'S

\* The data was obtained from measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-9.00 lens, 0.075mm center thickness).

<sup>1</sup>Lerman,S., Radiant Energyand the Eye, MacMillan, New York, 1980, p. 58, figure 2-21

<sup>2</sup>Waxler; M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

## **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays onto the retina.

The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

## INDICATIONS (USES)

ACUVUE OASY® Brand Conta¢ Lenses 1-Day with Hydraluxe<sub>TM</sub> Technology are indicated *tor* daily disposablewear *tor* the optical correction *ot* retracitveametropia (myopia and hyperopia)in phakic or aphakic persons with non-diseasedeyes who may have 1.00D or less *ot* astigmatism.

ACUVUE OASY® Brand Contact Lenses 1-Day with Hydraluxe<sub>TM</sub> Technology tor ASTIGMATISMare indicated *tor* daily disposable wear *tor* the optical correction *ot* refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-disease dyes who may have 0.50D to 3.00D *ot* astigmatism.

These lenses contain a UV Blocker to help protect againsttransmission *ot* harmtul UV radiationto the cornea and into the eye.

### CONTRAINDICATIONS (REASONS NOT TO USE)

# DO NOT USE these contact lenses when any of the following conditions exist:

- Acute or subacuteintlammationor intection ot the anterior chamber ot the eye.
- Any eye disease injury or abnormality that affects the cornea conjunctiva, or eyelids.
- Severe insufficiency ot lacrimal secretion (dry eye).

- Corneal hypoesthesia (reduced corneal sensitivity).
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocularirritation due to allergic reactions which may be caused by use of contact lenssolutions (i.e., rewetitng drops) that contain chemicalsor preservatives (such as mercury, Thimerosal, etc.) to which some people may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral).
- If eyes become red or irritated.

## **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEM\$, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLV AND LEAD TO LOSS OF VISION; IF THE PATIENT EXPERIENCES:

- Eye Discomfort,
- Excessive Tearing,
- Vision Changes,
- Loss of Vision,
- Eye Redness,
- Or Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY RE-MOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

 When prescribed for daily wear, patients should be instructed not to wear lenses while sleeping. Clinical studies have shown that the risk of serious adverse reactions is increased when lenses are worn overnight, and that the risk of ulcerative keratitis is greater for
extended wear contact lens users than for daily wear users3.

- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.
- The overall risk of ulcerativekeratitismay be reduced by carefully following directions for lens care.

#### **Specific Instructions for Use and Warnings:**

Water Activity

#### Instructions for Use

Do not expose contact lenses to water while wearing them.

#### **WARNING:**

Water can harbor microorganisms that can lead to severe infection vision lossor blindness of lenses have been submersed water when participating water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

### **PRECAUTIONS**

### **Special Precautions for Eye Care Professionals:**

• Due to the small number of patients enrolled in clinical investigation of lenses, ali refractive powers, design configuration, or lens parameters available in the lens materialare not evaluated in significant numbers. Consequent, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, centra! and peripheral thickness, and optic zone diameter.

<sup>&</sup>lt;sup>3</sup> New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

- The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.
- Patients who wear these lenses to correct presbyopia using monovision may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes. The lenses absorb this dye and become discolored.
   Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove the lenses immediately if the eyes become red or irritated.

# Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

### Handling Precautions:

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.
- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the "Patient Instruction Guide" for the prescribed

wearing schedule and those prescribed by the Eye Care Professional.

- Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container unless specifically indicated for that use. Slide the lens up the side of the bowl until it is free of the container.
- Do not touch the lens with fingernails.

### **Lens Wearing Precautions:**

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for a Sticking (Non-Moving) Lens." The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.
- The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hair spray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.
- Always discard lenses worn as prescribed by the Eye Care Professional.

#### **Lens Care Precautions:**

• The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

#### Other Topics to Discuss with Patients:

- Always contact the Eye Care Professionabefore using any medicine in the eyes.
- Certain medication, ssuch as antihistamine, sdecongestants, diuretics, muscle relaxants, tranquilizer, sand those for motion sickness may cause dryness of the eye, increased lens awareness, or blurredvision. Should such conditions exist, proper remedial measures should be prescribed. Depending on the severity, this could include the use of lubricating drops that are indicated for use with soft contact lenses or the temporary discontinuance of contact lenswear while such medication is being used.
- Oral contrace tive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- As with any contactlens, follow-up visits are necessary to assure the continuing health of the patient'seyes. The patient should be instructed as to a recommended follow-up schedule

### Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Profession as) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

### ADVERSE REACTIONS

# The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may bum, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to

# **Clinical Study Protocol**

CR-6501, v 4.0

peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis; some of which are clinically acceptable in low amounts.

- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows, or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be instructed NOT to use a new lens as self-treatment for the problem.

The patient should be advised that when any of the above symptoms occur, a serious condition such as intection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.


#### GENERAL FITTING GUIDELINES

#### A. Patient Selection

Patients selectedto wear these lenses should be chosen based on:

- · Motivation to wearlenses
- Ability to tollow instructions regarding lens wear care
- General health
- Abiilty to adequately handle andcare for thelenses
- · Ability to understand the risk and benefits of lens wear

Pa tients who do not meet the  ${\tt above}$  crtteria should not be provided with contact lenses.

#### B. Pre-fitting Examinatio

Initial evaluation of thepatientshould begin with a thorough casehistory to determinelf lhere are any contraindications to contactlenswear. During the casehistory, the patient svisual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preoeding the initial selection of trialoontact lenses, a comprehensive oblar evaluation shouldbe performed that includes, but is not limited to, the measurement of distance and near visual aculty, distance and near refractive prescription (including determining the preferred reacting distance tor presbyopes,) keratometry, and biomicroscopic evaluation.

Based on this evaluation, if It is determined that the patient Is eligible to wear these lenses, the Eye Care Professional should prooeed to the lens fitting instructions asout Ined below.

#### C. InItial Power Detennination

Aspectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance therefraction is greater than :t4.000.

#### D. Base Curve Selection (Trial Lens Fitting)

The following triallenses should be selected for patientsregardless of **kera**\* tometryreadings. However.oorneal curvature measurements shouldbe performed to establish the patient'sbasellneocular status.


- ACUVUE OASY\$1-Day: 8.5 mm/14.3 mm
- ACUVUE OASYS® 1-Day tor ASTIGMATISM: 8.5 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

### 1. Criteria of a Properly Fit Lens

Aproperly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

#### 2. Criteria of a Flat Fitting Lens

Aflat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink, and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

### 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

### E. FinalLens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.250 |
| Fina! lens power: | -2.25D |

| Example 2 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |
| Final lens power: | -1.750 |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see dispensing and follow up information in **PATIENT M ANAGEMENT**).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing ACUVUE OASYS® 1-Day for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the patient.

### A. How to Determine Lens Cylinder and Axis Orientation

#### 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm trom the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position - there is no "top" and "bottom" as ina prism-ballastedlens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.



You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

### 3. Assessing Rotation

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift", measure or estimate the "drift", then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.

#### B. Final Lens Power

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

### 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx  $> \pm 4.00$ D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx  $\leq \pm 4.00$ D, vertex compensation is not

necessary.

### 2. For the Cylinder

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq$  0.50D from the refractive cylinder.

### 3. Case Examples

### Example 1

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20 O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis 180°. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx Prescribed: O.D. -2.50D / -1.25D x 180° O.S. -2.00D / -0.75D x 180°

#### Example 2

Manifest (spectacle) refraction:

O.O. -3.00D *I* -1.00D x 90° 20/20

O.S. -4.75D *I* -2.00D x 90° 20/20

Choose diagnostic lenses of -3.00D / -0.75D x 90° for the right eye and -4.50D / -1.75D x 90° for the left eye, the nearest lenses available to the spherical power, cylinder power, and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

#### Right Eye

The orientation mark on the right lens rotates left from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx Prescribed: O.O.  $-3.00D I - 0.75D \times 100^{\circ}$ 

#### Left Eye

The orientation mark on the left lens rotates right from the 6 o'clock position by 10° and remains stable in this position.

Compensate for the 10° axis drift by subtracting it from the manifest refraction axis.

Here is the Rx Prescribed:

O.S. -4.50D I -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see dispensing and follow-up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### MONOVISION FITTING GUIDELINES

#### A. Patient Selection

#### 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.000) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot
  meet state driver's licensing requirements with monovision
  correction should be advised to not drive with this correction,
  OR may require that additional over-correction be prescribed.

#### 2. Patient Education

Ali patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu ina dim restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary tor the patient to realize the disadvantages as well as the advantages of clear near vision and straight ahead and upward gaze that monovision contact lenses provide.

#### **B.** Eye Selection

#### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1: Determine which eye is the "sighting eye." Havethe patientpoint to an object at the far end of the room.

Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting)eye.

Method 2: Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correcitonis in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

### 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### Refractive Error Method

For anisometropic correciton, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### Visual Demands Method

Conside the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

### C. Special Fitting Characteristics

#### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral myope would require correcitve lenses on

both eyes.

#### **Examples**:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the GENERAL FITTING GUIDELINES for base curve selection described in this Package Insert.

Case history and standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under

conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

### D. Other Suggestions

The success of the monovision technique may be further improved by having the patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Having supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Reftne the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clearnear vision and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

Ali patients should be supplied with a copy ot the PATIENT INSTRUCTION GUIDE tor these lenses. Copies are available tor download at www.acuvue.com.

### PATIENT MANAGEMENT

#### **Dispensing Visit**

Each sterile lensis supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. To remove the lens from the container, peel back the foil seal, place a finger on the lens, and slide the lens up the side of the bowl of the lens package until it is free of the container.

- Evaluate the physical fit and visual acuity of the lens on each eye.
- Teach the patient how to apply and remove his or her lenses.
- Explain daily disposable lens wear and schedule a follow-up examination.
- Previde the patient with a copy ot the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

#### Follow-Up Examinations

Follow-up care (necessary to ensure continued successful contact lens wear) should include routine periodic progress examinations, management of specific problems, if any, and a review with the patient of the wear schedule, daily disposable modality, and proper lens handling procedures.

# **Clinical Study Protocol**

CR-6501, v 4.0

Recommended Follow-up Examination Schedule (complications and specific problems should be managed on an individual patient basis):

- 1. One week from the initial lens dispensing to patient
- 2. One month post-dispensing
- 3. Every three to six months thereafter

**NOTE:** Preferably, at the follow-up visits, lenses should be worn for at least six hours.

#### Recommended Procedures for Follow-up Visits:

- 1. Solicit and record patient's symptoms, if any.
- Measure visual acuity monocularly and binocularly at distance and near with the contact lenses.
- Perform an over-refraction at distance and near to check for residual refractive error.
- With the biomicroscope, judge the lens fitting characteristics (as described in the GENERAL FITTING GUIDELINES) and evaluate the lens surface for deposits and damage.
- Following lens removal, examine the cornea and conjunctiva with the biomicroscope and fluorescein (unless contraindicated).
  - The presence of vertical corneal striae in the posterior central cornea and/or corneal neovascularization is indicative of excessive corneal edema.
  - The presence of corneal staining and/or limbal-conjunctival hyperemia can be indicative of an unclean lens, a reaction to solution preservatives, excessive lens wear and/or a poorly fitting lens.
  - Papillary conjunctival changes may be indicative of an unclean and/or damaged lens.
- Periodically perform keratometry and spectacle refractions. The values should be recorded and compared to the baseline measurements.

If any observations are abnormal, use professional judgment to alleviate the problem and restore the eye to optimal conditions. If

the criteria for successful fit are not satisfied during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

# WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to overwear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professionlabased upon the patient's physiological eye condition, because individua! response to contact lenses varies.

The maximum suggested wearing time for these lenses is:

| Day | Hours |
|-------------|-----------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | allwaking hours |

### REPLACEMENTSCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

### LENS CARE DIRECTIONS

When lenses are prescribed for daily disposable wear, the Eye Care Professional should provide the patient with appropriate and adequate warnings and instructions for daily disposable lens wear at the time they are dispensed

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have spare lenses or spectacles available.

#### Bas ic Instruct ions

- Always wash, rinse, and dry hands before handling contact lenses.
- Do not use saliva or anything other than the recommended solutions tor lubricating or rewetting lenses. Do not put lenses in the mouth.
- Eye Care Professionals may recommend a lubricating/rewetting solution which can be used to wet (lubricate) lenses while they are being worn to make them more comfortable.

#### Care for a Sticking (Non-Moving) Lens

If the lens sticks (stops moving), the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should immediately consult the Eye Care Professional.

### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISITAHOSPITAL EMERGENCY ROOM WITHOUT DELAY.

### **HOW SUPPLIED**

Each UV-blocking sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. The plastic package is marked with the following:

- ACUVUE OASYS® 1-Day:base curve, power, diameter, lot number, and expiration date
- ACUVUE OASYS® 1-Dayfor ASTIGMATISMbase curve, power, diameter, cylinder, axis, lot number, and expiraitondate

# REPORTING OF ADVERSE REACTIONS

Ali serious adverse experiences and adversereactionsobserved in patients wearing theselenses or experiencedwith these lensesshould be reported to:

Johnson& Johnson Vision Care, Ine. 7500 CenturionParkway Jacksonville, FL 32256 USA

Tel: 1-800 -843-2020 www.acuvue.com

CR-6501, v 4.0

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA

Tel: 1-800-843-2020 **www.acuvue.com** 



©Johnson & Johnson Vision Care Companies 2016 In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed in USA.

> Revision date: 09/16 Revision number: AO-03-16-13

ACUVUE OASYS® and HydraLuxe™ are Trademarks of the Johnson & Johnson Vision Care Companies

# APPENDIX D:

- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL
  REFRACTIVE ERROR
- BIOMICROSCOPY SCALE
- DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION



Lens Fitting Characteristics Title: Document Type: **Document Number:** Revision Number: 6

Lens Fitting Characteristics Title: Document Type: **Document Number:** Revision Number: 6

CR-6501, v 4.0 JJVCCONFIDENTIAL Page 131 of160

Lens Fitting Characteristics Title: Document Type: **Document Number:** Revision Number: 6

#### Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Lens Fitting Characteristics

Title: Lens Fitting Characteristics

Document Type:

Document Number: Revision Number: 6



**Clinical Study Protocol** 

| Johnson & Johnson Vision | Care, Ine. |
|-------------------------------------|--------------------|
| Title: Lens Fitting Characteristics | ,<br> |
| Document Type: | |
| Document Number: | Revision Number: 6 |
| Document Number: | Revision Tumber. 0 |

CR-6501, v 4.0



Clinical Stud y Prntocol Johnson & Johnson Vision Care, Ine. Title-----Subject Reported Ocular Symptoms/Problems

Document Type: Document Number: Revision Number: 4


DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS





# **Clinical Study Protocol**

Johnson & Johnson Vision Care, Inc. Determination of Distance Spherocylindrical Refractive Error

Title: Determination of Distance Spherocylindrical Re
Document Type:

Document Number: Revision Number: 5

Title------ Determination of Distance Spherocylindrical Refractive Enor Document Type: **Document Number: Revision Number:** 5

Title------ Determination of Distance Spherocylindrical Refractive Enor Document Type: Document Number: **Revision Number:** 5

Title------ Determination of Distance Spherocylindrical Refractive Enor Document Type: Document Number: **Revision Number:** 5






Title: **Biomicroscopy Scale** DocumentT ype: Revision Number: 10 **Document Number:** 


Title: **Biomicroscopy Scale** DocumentT ype: Revision Number: 10 **Document Number:** 


Title: **Biomicroscopy Scale** DocumentT ype: Revision Number: 10 **Document Number:** 


| litle: | Blomicroscopy Scale | |
|------------------|---------------------|---------------------|
| Document Type: | | |
| Document Number: | | Revision Number: 10 |
| 2 | | |
| _ | | |
| | _ | |
| I | | |
| I | | |
| | | - |



Title----- Distance and Near Snellen Visual Acuity Evaluation Document Type: Revision Number: 5 **Document Number:** 



Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Distance and Near Snellen Visual Acuity Evaluation

Title:

**Document Type: Document Number: Revision Number: 5** 

Title----- Distance and Near Snellen Visual Acuity Evaluation
Document Type: Document Number: **Revision Number: 5** 

Title----- Distance and Near Snellen Visual Acuity Evaluation

Document Type: **Document Number:** Revision Number: 5




APPENDIX E: GUIDELINES FOR COVID-19 RISK MITIGATION

| _Title Guidelines for | COVID-19Risk Mitigation |
|-----------------------|-------------------------|
| Document Ty e: | |
| Document Number: | Revision Number: 5 |

#### 1.0 PURPOSE

The purpose of this document is to provide guidelines for the re-opening or initiation of clinical study sites participating in Johnson & Johnson Vision Care, Inc. (JJVCI) clinical studies during the COVID-19 pandemic.

#### 2.0 SCOPE

This document provides guidelines for Johnson & Johnson Vision Care (JJVCI) to address the potential risks from COVID-19 to study subjects, investigators, study site staff, and monitors at study sites. The guidance provided in this document is in effect from the date of approval through the date of retirement of this Work Instruction. At a minimum, this Work Instruction will be reviewed and updated on a quarterly basis, as appropriate.

NOTE: Re-opening of sites outside of the US will be evaluated on a country by country basis subject to local health authority guidance.

#### 3.0 **DEFINITIONS**

American Academy of Optometry (AAO): The American Academy of Optometiy is an organization of optometrists based in Orlando, Florida. Its goal isto maintain and enhance excellence in optometric practice, by both promoting research and the dissemination of knowledge. The AAO holds an annual meeting, publishes a monthly scientific journal, gives credentials to optometi-ists through the fellowship process and publishes position statements.

American Optometric Association (AOA): The American Optometl'ic Association, founded in 1898, is the leading authority on quality care and an advocate for our nation's health, representing more than 44,000 Doctors of Optometry (O.D.), optometric professionals, and optometry students. Doctor of Optometry take a leading role in patient care with respect to eye and visi011care, as well as general health and well-being. As primary health care providers, Doctor of Optometry have extensive, ongoing training to examine, diagnose, treat and manage ocular disorders, diseases and injuries and systemic diseases that manifest in the eye. The American Optometric Association is a fe.deration of state, student, and anned forces optometic associations. Through these affiliations, the AOA serves members consisting of optometi'ists, students of optometry, paraoptometicicassistants and technicians. The AOA and its affiliates work to provide the public with quality visi011and eye care.

Centers fo1 Disease Control and Prevention (CDC): The Centers for Disease Control and Prevention is a national public health institute in the United States. It is a United States federa! agency, under the Department of Health and Human Services, and is headquartered in Atlanta, Georgia.

**COVID-19:** CtuTent outbreak of respiratory disease caused by a nove! coronavirus. The virus has been named "SARS-CoV-2" and the disease it causes has been named "Coronavirus Disease 2019" (COVID-19).

Clinical Study: Volw1taiyresearch studies conducted in people and designed to answer specific questions about the safety or effectiveness of drugs, vaccines, other therapies, or new ways of using existing ti-eatinenst. May also be called clinical trials, studies, research, ti-iasl, or protocols.

Clinical Study Site: Location where a clinical study is conducted, such as a doctor's office, university, or laboratory. Clinical studies are conducted by Investigators who are individual(s) responsible for the conduct of the clinical study at a study site. If a study is conducted by a team of individuals, the Investigator is the responsible leader of the team and may be called the Principal Investigator.

**Clinical Operations Manager (COM):** The Johnson & Johnson Vision Care (JJVCI) individua! responsible for the overall management of a clinical trial.


| <u> 11016</u> | Guidennes for <u>CC</u> | V ID-19 KISK MIUSauon | |
|---|---|---|---|
| Document Ty e: | | | |
| Document Number: | | R | evision Number: 5 |

**Monitor:** An individua! designated to oversee the progress of a clinical study and ensure that it is conducted, recorded, and repolted in accordance with the protocol, Standard Operating Procedures (SOPs), Good Clinical Practice (GCP), and applicable regulat01y requirements.

Medical Safety Office1 (MSO): Physician who has primally accountability in their product polltfolio for product health and safety, and who serves as an independent medica! voice for patient safety.

**Safety Management Team (SMT):** A cross-functional, collaborative team responsible for review, assessment and evaluation of medica! safety data arising from any source throughout the product life cycle.

#### 4.0 GUIDANCE FOR STUDY DOCUMENTS

In alignment with recent health authority guidance, JNCI is providing recommendations for study-related management in the event of dismption to the conduct of the clinical study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health, safety and well-being of palticipants and site staff. If, at any time, a palticipant's safety is considered to be at risk, study intervention will be discontinued, and study follow-up will be conducted as outlined in the protocol.

During the COVID-19 pandemic, the additional risks listed below need to be considered for study pa1 ticipants and study personnel:

#### 4. I Additional Risks Related to the COVID-19 Pandemic:

- The possible transmission of the Coronavims infection and consequent complications, beyond the risk of adverse events due to the investigational device and/or procedures.
- The risk may be higher in an optometric clinical study because of the close contact the subject will have with heaith care professionals dwing the procedures and assessments (since the investigator must make the measwements close to the subject's face) and, in addition the need for multiple follow-up visits/exams which may expose the subject to other patients and/or healthcare professionals who might be transmitting the vims, even if they do not have symptoms.
- Potential dismptions to the study may be necessaly due to cun-ent or future pandemic-related emergency restrictions, which may lead to delays in scheduled follow-up visits.
- Subjects experiencing an adverse event related to contact lens wear may receive delayed treatment
  due to COVID-19 restrictions. 1nthis event, all assessments that can be conducted virtuaUy will be
  completed by the investigator to detennine the best course oftreatment for the subject, including
  an unscheduled visit, up to discontinuation from the study, as appropriate.

If a study subject is found to have contracted COVID-19 during palticipation in a study, he/she will be discontinued from the study and followed until COVID-19 Adverse Event (AE) resolution.

To help minimize the above potential risks, JNCI recommend reviewing/complying with local, state, and governmental guidance for COVID-19 risks.

JNCI will provide the following studyspecific documents with language peltaining to COVID-19 risks:

#### 4.1.1 Info1med Consent:

Will include info1mation concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Infonned Consent document:

Page 2 of ll

| <u>Title</u> | Guidelines for <u>CC</u> | OVID-19Risk Mitigation | |
|---|---|---|---|
| Do cument Ty e: | | | |
| Document Number: | 7 | | Revision Number: 5 |

#### STUDY ASSOCIATED RISKS RELATED TO COVID-19 (CORONAVIRUS) PANDEMIC

It is important to note that this study will be conducted, at least in pali, during the COVID 19 pandemic. As such, additional risks associated with the infection with COVID-19 exist for you. This is palticularly important for this study due, in part, to the closeness of the doctor during the study examinations.

The potential effects of the disease are not fully known, at this time, and may include long-tenn serious health consequences. In severe cases, this may result in hospitalization and/or death. Based on ctment knowledge from the Centers for Disease Control and Prevention (CDC), those at high-risk for severe illh1ess from COVID-19 include older adults and people with underlying medica! conditions.

During this study, all appropriate measures will be taken to minimize risks including the use of personal protective equipment such as masks and gloves, as well as proper sanitization. This is in conf01mance to guidance from the CDC, local health deprut ments, and the state and county in which the study doctor's office is located. However, these measures may not completely eliminate the risks associated with contracting COVID-19.

Ifyou ru e found to have contracted COVID-19 or feel ill with flu-like symptoms during participation in the study, you will not be pel mitted to continue in-office study follow-up visits, but you will receive instructions and your condition will be monitored by the doctor and/or study staff.

#### 4.1.2 COVID-19 Risk Control Checklist (Attaclunen-tB):

Will include COVID-19 risk control methods that are required by a site to conduct JNCI clinical studies. The risk controls are consistent with CDC, AOA, AAO Guidance. The Principal Investigator will review/sign the study specific checklist prior to the Site Initiation Meeting.

#### 4.1.3 Protocol Compliance Investigato(rs) Signature Page:

Will include a statement indicating that the Principal Investigator (PI) agrees to conduct the study in compliance with all local, state, and govenuental guidance's for COVID-19 risk mitigation.

I have read the suggested guidance provided by JNCI pertaining to the COVID-19 risk mitigation, (COVID-19Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, govenunental guidance for COVID-19 risks.

#### 4.1.4 Study Site Initiation Training Slides:

Will include suggestions to help mitigate potential transmission of COVID-19. Suggestions may include maintaining social distancing in the clinical site by staggered scheduling of study patients, wearing proper PPEs, frequent disinfection, and installing shields on the slit lamp and other applicable equipment.

#### S.O **GUIDANCE FOR REMOTE SUBJECT VISITS**

Potential dismptions to the study may be necessary due to cmTent or future pandemic-related emergency restrictions. Possible disruption of the study as a result of COVID-19 control measures may lead to delays in scheduled follow-upvisits.

Subjects may be delayed in being seen for study follow up visit(s), for exrunple due to COVID-19 control measures or due to the subject's concems or fears about COVID-19 risk. When appropriate, the remote assessment will be conducted to the extent possible. Discussions with the subject during remote assessments may include:


| <u> 11tle</u> | - Guidelines for <u>CC</u> | DVID-19 Risk Mitigation | |
|---|---|---|---|
| <b>Document Ty e:</b> | | | |
| Document Number | | _ | Revision Number: 5 |

| Procedure | Details |
|---|---|
| Subject Repo1ted Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire regarding the test article when applicable and feasible. |
| Change of Medical History<br>(Adverse Events) and<br>Concomitant Medications /<br>Therapies Review | Record any adverse events or medical history changes from the previous study visit with the subject/parents. Review the subject's concomitant medications/therapies and record any changes from the previous study visit. |
| Wearing Time and Compliance | Record the a:verage wearing time (including number ofhow-s per day during weekdays and weekends, and number of days per week). Confinn compliance with the prescribed wear schedule. Record and discuss the lens wear compliance based on the subject's self-repolt. For example, the subjects will be a.sked the time of the day the subject typically puts on the study lenses in the moming and takes off in the evening, the number of days per week lenses were wom, and the mllllber of consecutive days the subject didn't wear the study lenses, etc. |

The discussion with the subject will be documented in EDC under Tele-Visit and a minor protocol deviation will be noted. If during the telephone consultation, a subject states he/she wishes to discontinue participating in the study, instruct the subject to stop wearing the study lenses and schedule the subject to return to the clinic for a Final Evaluation at the at earliest possible time. Subjects should return all wmsed lenses to the clinic at the la.st visit.

Changes in study visit schedules, missed visits, or participant discontinuations may lead to missing data, including data related to protocol-specified procedures. Case repolt fonns should capture specific infolmation regarding the basis of missing data, including the relationship to the COVID-19 pandemic.

#### 6.0 STUDY CONDUCT DURINGPANDEMIC

It is recognized that the Coronavims Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantineby participants and study-site personnel; trave! rest1·ictions/lin1ited access to public places, including Optometly Clinics; and changes in clinic procedures required to address the COVID-19 challenge.

Evely effort should be made to adhere to protocol-specified assessments for study participants, including follow-up. However, if scheduled visits cannot be conducted in person at the study site it is suggested that assessments be pelfolm ed to the extent possible remotely/vit1ually or delayed wltil such time that on-site visits can be resumed it1 order to continue pruticipant monitoring in a.ccordat1ce with the protocol where possible. At each contact, pru-ticipants will be it1terviewed to collect safety data. Key effica.cy endpoit1t assessments should be perfolmed if required ruld as feasible.

Modifica.tions to protocol-required assessments may be pennitted via COVID-19 Appendix after consultation with the prut icipant, itiv estigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol devia.tions. Inten uptions of test ruticle wear or discontinuations of study it1terventions and withdrawal from the study should be documented with the prefix "COVID-19-related" it1 the ca.se report f01m (CRF).


| <u> 1 1t1e</u> | Guidelines for <u>CC</u> | VID-19 RISK WIITIGATION | |
|---|---|---|---|
| Document Ty e: | | | |
| Document Number: | | Revi | sion Number: 5 |

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance.

If a patticipant has tested positive for COVID-19, the investigator should contact the sponsor's responsible medical monitor to discuss initial plans for study intervention and follow-up. The medical monitor will notify the Safety Management Team of any subject(s) that have repolted "COVI D-19", "Asymptomatic COVID-19", or "S uspected COVID-19" adverse events within 24 hours of the notification.

Modifications made to the study conduct as a result of the COVID-19 pandemic will be summarized in the clinical study repolt.

COVID -19 scr eening procedures that may be mandated by local healthcare systems do not need to be repolted as an amendment to the protocol even if done during clinical study visits.

#### **6.1** Monitoring Visits

When on-site monitoring by the sponsor is not feasible, the sponsor's site monitor will contact the study site to schedule remote visits. In such cases, on-site monitoring visits will resume when feasible, with increased frequency to address the source data verification backlog.

Even with staffing linitations during this COVID-19 pandemic, aU routine operations related to clinical trials should be well-documented and at chived as part of standard process. When conditions permit, all pruties involved in this clinical trial should communicate relevant information in a timely manner so that all relevant parties remain sufficiently infol med.

#### 6.1.1 Study Site Initiation:



On-site visits may be considered when, for example, hands-on training or evaluation of site facilities is required. While on site, the Clinical Research Associate (CRA) will follow aU local, stat e, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

#### 6.1.2 Interim Monitoring Visits (if applicable):

During the period that this Work Instruction is in effect, Interim Monitoring On-site visits will be kept to a minimum and include only those tasks that the CRA cannot pelform remotely (e.g., source document verification, test alticle reconciliation, etc.).

To ensur e data integrity during the conduct of ali JJVC studies, clinical study teams will follow the study specific Clinical Monitoring Plan

While on site, the CRA will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, weating of PPE, etc. as applicable for the location of fue study site.

Page 5 of II


Page 5 of ll


Title: Guidelines for CO VI D rus 9k Mir ati o n

Document Ty e:

Document Number:

Revision Number: 5

#### 6.1.3 Study Site Closure:

During the period that this Work Instn1ction is in effect, the duration of the Study Site Closure Visit will be limited to tasks that the CRA cannot perfonn remotely (e.g., sow ce document verification, test article final reconciliation and retw1,1etc.).


| Title Guidelines for | COVID-19Risk Mitigation |
|----------------------|-------------------------|
| Document Ty e: | |
| Document Number: | Revision Number: 5 |

At tachment A: Stud y Site Col'l'espondence

XXXX XX, 2020

#### Re: COVID-19 Mitigation Plan, << CR-xxxx/protocol title>>

Dear << Principal Investigator>> and Study Team,

Coronavirns (COVID·19) has impacted several conununities and business activities over the past several months. While we work toward the successful conduct of clinical studies, our conunitment continues to be the safety of patients, healthcare professionals, and to om conununities.

Therefore, we would like to share the following revisions/additions related to the above referenced Johnson & Johnson Visi011Care company sponsored clinical trial(s) you are etmently working on or considering palticipation within.

#### **Protocol:**

• Guidelines for COVID-19 Risk Mitigation provided in the Appendix section.

#### **Protocol Signature Page:**

 Will include a sta. tement indicating the Principa. I Investigator agrees to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

#### **Informed Consent:**

• Will include infonnation concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Infonned consent document.

#### COVID-19 Risk Control Checklist fot Clinical Studies:

• Will include COVID-19 risk control mea.sme s that are required to ensme the safety and health of subjects, site staff and monitors during the pandemic.

We want to encourage the need for open lines of communication a bout potential challenge s you may foresee as the result of the cun-ent COVID-19 situation. Therefore, we encourage you to regularly connect with your respective Johnson & Johnson clinical study team (Clinical Research Associate (CRA), Lead CRA or Study Managers).

Thank you for your continued engagement, collaboration, and dedication to your study subjects during this challenging time.

Please file this letter in your site file study con-es pondence.

Pag e 171 of 160


| <u>_Title</u> | - Guidelines for <u>CC</u> | OVID-19Risk Mitigation | |
|---|---|---|---|
| <b>Document Ty e:</b> | | | |
| <b>Document Number:</b> | | | Revision Number: 5 |

#### Attachment B: COVID-19 Risk Control Checklist

Study Number Site Number Principal Investigator (PI) Name

The followi.ng COVID -19 risk co.ntrol methods ru $\cdot$ e required to co.nduct Johnso.n & Johnso.n Vison Cru $\cdot$ e cli.nical studies . Plea se review the follo wi.ng requirements a.nd I.nitial each requirement.

| PI Initials | General Site Safety PlannirnzMeasures |
|---|---|
| | Silmaize w ith i.n s ite de s cribin iz Ri s k Control methods |
| | Social Distanci.niz oractices throughout site (waiti.niz room s lobby, exam rooms, etc.) |
| | Non-contact thermometer available to assess temoeratures of staff ruld on tient s |
| | Trai.niniz on oatient flow and ohvsical distanci.niz i.n waiti.niz room |
| | Establish lonizer time frame between oatient annointments to reduce oersons i.n the s ite |
| | Staff should receive job-specific traini.ng on PPE and demon strate compe tency with selection a.nd proper use of PPE ruld wear at ali times during i.nteraction s with subjects (e.g., putting on and removing without self-contami.nation) |

| P I Initials | Site Staff Daily Safety Measures |
|---|---|
| | As part of routine practic.e, si te staff should regularly monitor themselves for fever and symptoms of COVID-19 i.ncludi.ng temperature checks |
| | A.ny staff member (including 11011s-tudy clinic staff and Investigators) showi.ng s igns ofbei.ng sick or testing positive for COVID-19 must not be pennitted to work on activity that may expose study related staff ru1d subject and the Sponsor shall be i.nformed NOTE: Inform JJVC in 24 how·s of any COVID-19 cases and all potentfal exposure dw'ing the dinical study. |
| | Ensure that all staff wear a mask Gloves should be reauired when working directly with oatients ruld changed between each oatient |
| | Have staff thoroughly wash hands for at least 20 seconds or use rul a lcohol-ba s ed hruld s anitizer when they ruri ve. before and after each oatient before eating and aBer using the bathroom. |
| | Cleru1i.ng ru1d disi.nfection procedure s for exrun rooms and instruments or equipment between oatients with izlo v e s . |
| | Cleru1i.ng ru1d disinfection procedures for collllllonly touched surfaces (doors, chairs, computers, phones, etc.) with gloves. |

| PI Initials | Before a Patient or Study Visit: |
|---|---|
| | Patients should be asked prior to enteri.ng the site about fever and respiratory illness and whether they or a frunily member have had contact with another person with confinned COVID-19 i.n the past 14 days. Patients exhibiting signs ofbei.ng sick should be rescheduled when their symptoms resolve. |
| | Instruct patients that companions should remain outside of the facility ruld not accompany the patient i.nto the facility unless they are a parent/guardianof the patient or if they rue a trne cruegiver and need to assist the oatient |
| | Request the patient to call or text the office upon all'ival so entrance to and movement through facility can be coordi.nated by site staff |


| <u>litle</u> | Guidelines for <u>CC</u> | DVID-19Risk Mitigation |
|------------------|--------------------------|------------------------|
| Document Ty e: | | |
| Document Number: | | Revision Number: 5 |

| PI Initials | Patients Entering the site: |
|---|---|
| | Temperatme checks utilizing a non-contact thennometer for ali patients and companions entering the site. |
| | Alpi atien ts and companions must wear cloth or disposable mask at all times in the site |
| | Maintain social distancing. Waiting rooms or lobbies should be as empty as possible. Advise seated patients to remain at least 6 feet from one another. |
| | Communal objects in (e.g. toys, reading materials, etc.) should be removed or cleaned re larly. |

I certify that I have read and agree to implement ali the listed COVID-19 Risk Control Measures required for the conduct of Johnson & Johnson Visi011Care studies.

Principal Investigator Signature and Date


| <u>Title</u> | - Guidelines for <u>CC</u> | OVID-19Risk Mitigation | |
|---|---|---|---|
| Document Ty e: | | | |
| Document Number: | | | Revision Number: 5 |

Title ----- Guidelines for COVID-19Risk Mitigation

Document Ty e:

Document Number:

Revision Number: 5

#### RESOURCE LINKS

#### **US Resource Links**

OSHA Training

https://www.osha.gov/SLTC/covid-19/controlprevention.html

Personal Protective Equipment (PPE) Training

CDC: https://www.cdc.gov/coronavims/2019-ncov/hcp/using-ppe.html

I&R Training

ACUVUE® Len sA ss ist: http s://www.acuvue.com/lensassist

• Clinic Preparedness Guides

CDC: https://www.cdc.gov/coronavinis/2019-ncov/hcp/clinic-preparedness html

AOA: <a href="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-guidance-for-re-opening-practices-covid-19/1?m4="https://aoa-guidance-for-re-opening-practices-guidance-for-re-opening-practices-guidance-for-re-opening-g

American Optometric Association: <a href="https://www.aoa.org/optometzy-practice-reactivation-prw.aredness-imide">https://www.aoa.org/optometzy-practice-reactivation-prw.aredness-imide</a>

lu-Office Disinfection of Multi-Patient Use Diagnostic Contact Lenses
 https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf

#### **OUS Resource Links**

- Updates on local regulations in Hong Kong\_ https://www.coronavims.govhk/eng/index.html
- Resumption of optical services in England: Letter from Matt Neligan and Poonam Shanna <a href="https://www.england.nhs.uk/coronavims/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf">https://www.england.nhs.uk/coronavims/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf</a>
- NHS Optical Letter
   <a href="https://www.englandnhs.uk/coronavims/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf">https://www.englandnhs.uk/coronavims/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf</a>
- The College of Optometrists primacy eye care COVID-19 guidance: Red phase
   https://www.college-optometrists.org/the-college/media-hub/news-listgi/ncoronavims-covid-19-guidance-for-optometrists.html
- The College of Optometrists COVID-19: College updates
   <a href="https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavims-2019-advice-for-optometrists.html#CollegeGuidelines">https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavims-2019-advice-for-optometrists.html#CollegeGuidelines</a>
- Infection Control Guidelines. (n.d.). Ret,rieved from Canadian Association Of Optometrists: https://opto.ca/sites/default/files/resources/documents/infection control gnidelines 2016.pdf
- Infection prevention and control for COVID-19: Interim guidance for outpatient and ambulato1y care settings. (2020, May 23 May). Retrieved from Government of Canada: https://www.canada.ca/en/public-health/services/diseases/2019-novel-coronavims-infection/guidance-documents/interim-guidance-outpatient-ambulato1ycare-settings html

Page 10 ofll

| Title Guidelines fo | · COVID-19Risk Mitigation |
|---------------------|---------------------------|
| Document Ty e: | |
| Document Number: | Revision Number: 5 |

- Info1mation for Members On Coronavirus (COVID-19). (n.d.). Retrieved from Canadian Association Of Optometrists:
  - https://opto.ca/sites/default/files/resources/documents/info1mation for members on coronavims.pdf
- Coronavirns (COVID-19) resources for health professionals, including aged care providers, pathology providers and health care managers. (2020, September 24). Retrieved from Australian Govennment Department of Health:
  - https://www.health.gov.au/resources/collections/coronavims-covid-19-resources-for-health-professionalsincluding-aged-care-providers-pathology-providers-and-health-care-managers
- Environmental Cleaning and Disinfection Principles for COVID-19. (n.d.). Retrieved from Australian Government Depallment of Health: https://www.health.gov.au/sites/default/files/documents/2020/03/environmental-cleaning-and-disinfectionprinciples-for-covid-19.pdf
- Infection control guidelines and advice. (11.d.). Re trie v ed from Optometiy Australia: https://www.optometiy.org.au/practice-professional-suppo1/coronavims-covid-19-what-optometrists-needto-know/covid-19-clinical-advice/infection -con ti-ol-guidelines-and-advice/

Page 11 ofll


#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6501 Protocol Title: Role of glare and spectral filtering on contrast sensitivity: A pilot study

Version and Date: 4.0 02 November 2022

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155:2020,<sup>1</sup> the Declaration of Helsinki,<sup>2</sup> United States (US) Code of Federal Regulations (CFR),<sup>3</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix E of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |